CLINICAL TRIAL: NCT03781167
Title: A 52-Week, Open-label, Single-arm Study to Evaluate the Safety and Tolerability of 24-hour Daily Exposure of Continuous Subcutaneous Infusion of ABBV-951 in Subjects With Parkinson's Disease
Brief Title: A Study to Evaluate the Safety and Tolerability of ABBV-951 in Subjects With Parkinson's Disease (PD)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M15-741; 2018-002144-85 (EudraCT Number)
Record Dates: First submitted 2018-12-18; First posted 2018-12-19 (Actual); Results first posted 2023-10-23 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-09

CONDITIONS: Parkinson's Disease (PD)
Keywords: Parkinson's Disease (PD); ABBV-951; Levodopa/Carbidopa
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- ABBV-951 Low Dose Subgroup (Experimental): After a 4-week Optimization Period, participants continued receiving ABBV-951 by continuous subcutaneous infusion (CSCI) during the 48-week Maintenance Period. Participants whose modal total daily dose (most frequent dose) over the entire study was < 2530 mg of Foslevodopa/day were analyzed as the Low Dose Subgroup.
  Interventions: Drug: ABBV-951
- ABBV-951 High Dose Subgroup (Experimental): After a 4-week Optimization Period, participants continued receiving ABBV-951 by continuous subcutaneous infusion (CSCI) during the 48-week Maintenance Period. Participants whose modal total daily dose (most frequent dose) over the entire study was ≥ 2530 mg of Foslevodopa/day were analyzed as the High Dose Subgroup.
  Interventions: Drug: ABBV-951

INTERVENTIONS:
Drug: ABBV-951 — Solution for continuous subcutaneous infusion (CSCI)
  Other Names: Foslevodopa/Foscarbidopa

SUMMARY:
The purpose of this study was to assess the safety and tolerability of ABBV-951 (Foslevodopa/Foscarbidopa) in participants with Parkinson's disease (PD).

This was a single-arm study with preplanned analyses conducted by dose subgroup (Low Dose or High Dose) based on the modal total daily dose (most frequent dose) over the treatment period.

ELIGIBILITY:
Inclusion Criteria:

* Participants with diagnosis of idiopathic Parkinson's Disease (PD) that is levodopa-responsive
* Participants must be judged by the investigator to be inadequately controlled by current therapy, have recognizable/identifiable "Off" and "On" states (motor fluctuations), and have a minimum of 2.5 hours of "Off" time per day

Exclusion Criteria:

* Participant is cognitively impaired and is not able to safely and effectively manage the drug delivery system and the diaries and is not able to adhere to the study
* Participant is considered by the investigator to be an unsuitable candidate to receive ABBV-951 for any reason

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 244 (Actual)
Dates: Start 2019-04-29 (Actual); Primary Completion 2022-08-17 (Actual); Study Completion 2022-08-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (65):
- United States (24):
  - University of Alabama at Birmingham - Main /ID# 207996, Birmingham, Alabama
  - Banner Sun Health Res Inst /ID# 208811, Sun City, Arizona
  - The Parkinson's & Movement Disorder Institute - Fountain Valley /ID# 216126, Fountain Valley, California
  - University of Colorado Hospital /ID# 207968, Aurora, Colorado
  - Parkinson's Disease and Movement Disorders Center of Boca Raton /ID# 207677, Boca Raton, Florida
  - Northwestern University Feinberg School of Medicine /ID# 208812, Chicago, Illinois
  - Indiana Clinical Research Cent /ID# 207952, Indianapolis, Indiana
  - Univ Kansas Med Ctr /ID# 208963, Kansas City, Kansas
  - University of Kentucky Chandler Medical Center /ID# 207603, Lexington, Kentucky
  - Massachusetts General Hospital /ID# 207993, Boston, Massachusetts
  - Health Partners /ID# 207950, Saint Paul, Minnesota
  - University of Missouri /ID# 209043, Columbia, Missouri
  - Washington University-School of Medicine /ID# 207525, St Louis, Missouri
  - Dartmouth-Hitchcock Medical Center /ID# 207972, Lebanon, New Hampshire
  - Wake Radiology UNC REX Healthcare - Raleigh Office /ID# 209784, Raleigh, North Carolina
  - Legacy Medical Group - Neurology /ID# 208031, Portland, Oregon
  - Prisma Health Cancer Institute-Faris Road /ID# 207650, Greenville, South Carolina
  - Neurology Consultants of Dallas - LBJ Fwy /ID# 207619, Dallas, Texas
  - Baylor College of Medicine /ID# 207620, Houston, Texas
  - Central Texas Neurology Consul /ID# 216918, Round Rock, Texas
  - Univ Texas HSC San Antonio /ID# 208958, San Antonio, Texas
  - Booth Gardner Parkinson's Care Center /ID# 208026, Kirkland, Washington
  - Inland Northwest Research /ID# 208122, Spokane, Washington
  - Medical College of Wisconsin /ID# 207999, Milwaukee, Wisconsin
- Australia (5):
  - Concord Repatriation General Hospital /ID# 207628, Concord, New South Wales
  - Westmead Hospital /ID# 207633, Westmead, New South Wales
  - Royal Adelaide Hospital /ID# 207634, Adelaide, South Australia
  - Alfred Health /ID# 207632, Melbourne, Victoria
  - Perron Institute /ID# 207627, Nedlands, Western Australia
- Belgium (3):
  - Universitair Ziekenhuis Leuven /ID# 209058, Leuven, Vlaams-Brabant
  - AZ Sint-Jan Brugge /ID# 208178, Bruges
  - Groupe Sante CHC - Clinique du MontLegia /ID# 208177, Liège
- Canada (2):
  - University of Calgary - Movement Disorders Clinic /ID# 207342, Calgary, Alberta
  - Centre de Recherche St-Louis /ID# 207344, Québec, Quebec
- Denmark (3):
  - Bispebjerg and Frederiksberg Hospital /ID# 207669, Copenhagen NV, Capital Region
  - Aarhus University Hospital /ID# 207668, Aarhus N, Central Jutland
  - Odense University Hospital /ID# 207871, Odense C, Region Syddanmark
- Germany (3):
  - Universitaetsklinikum Ulm /ID# 208602, Ulm, Baden-Wurttemberg
  - Kliniken Beelitz GmbH /ID# 208600, Beelitz-Heilstätten
  - InnKlinikum Haag /ID# 208601, Haag
- Italy (3):
  - IRCCS Centro Neurolesi Bonino Pulejo /ID# 207975, Messina
  - Fondazione IRCCS Istituto Neurologico Carlo Besta /ID# 207955, Milan
  - Azienda Ospedaliera di Padova /ID# 208077, Padua
- Japan (5):
  - National Hospital Organization Asahikawa Medical Center /ID# 210914, Asahikawa-shi, Hokkaido
  - National Hospital Organization Utano National Hospital /ID# 210912, Kyoto, Kyoto
  - Osaka University Hospital /ID# 210913, Suita-shi, Osaka
  - Juntendo University Hospital /ID# 210915, Bunkyo-ku, Tokyo
  - National Center of Neurology and Psychiatry /ID# 210911, Kodaira-shi, Tokyo
- Netherlands (2):
  - Erasmus Medisch Centrum /ID# 208168, Rotterdam, South Holland
  - St. Antonius Ziekenhuis /ID# 208529, Nieuwegein
- Russia (2):
  - Academician I.P. Pavlov First St. Petersburg State Medical University /ID# 216303, Saint Petersburg, Sankt-Peterburg
  - City Clinical Hospital #40 /ID# 216301, Sestroretsk, Sankt-Peterburg
- Spain (7):
  - Hospital General Universitario de Elche /ID# 209777, Elche, Alicante
  - Hospital Universitario de Bellvitge /ID# 209539, L'Hospitalet de Llobregat, Barcelona
  - Hospital Universitario A Coruna - CHUAC /ID# 212147, A Coruña
  - Hospital Santa Creu i Sant Pau /ID# 208240, Barcelona
  - Hospital Universitario Virgen de las Nieves /ID# 208242, Granada
  - Hospital Universitario Ramon y Cajal /ID# 208241, Madrid
  - Hospital Universitario Virgen del Rocio /ID# 208239, Seville
- Sweden (3):
  - Skane University Hospital Lund /ID# 207811, Lund, Skåne County
  - Centrum for neurologi /ID# 207716, Stockholm, Stockholm County
  - Sahlgrenska University Hospital /ID# 207718, Gothenburg, Västra Götaland County
- United Kingdom (3):
  - NHS Tayside /ID# 209242, Dundee, Scotland
  - King's College Hospital NHS Foundation Trust /ID# 208413, London
  - University Hospital Plymouth NHS Trust /ID# 208447, Plymouth

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible data sharing regarding the clinical trials we sponsor. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information (e.g., protocols, analyses plans, clinical study reports), as long as the trials are not part of an ongoing or planned regulatory submission. This includes requests for clinical trial data for unlicensed products and indications.
Time Frame: For details on when studies are available for sharing visit https://vivli.org/ourmember/abbvie/
Access Criteria: Access to this clinical trial data can be requested by any qualified researchers who engage in rigorous independent scientific research, and will be provided following review and approval of a research proposal and statistical analysis plan and execution of a data sharing statement. Data requests can be submitted at any time after approval in the US and/or EU and a primary manuscript is accepted for publication. For more information on the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- [Derived] Pahwa R, Aldred J, Soileau MJ, Standaert DG, Fung VSC, Kimber T, Malaty IA, Santos-Garcia D, Carroll C, Henriksen T, Parab A, Yan CH, Facheris MF, Spiegel A, Harmer L, Zamudio J, Chaudhuri KR. Improvement in Motor Consistency and Stability with Foslevodopa/Foscarbidopa in Advanced Parkinson's Disease: Post Hoc Analysis of Two Phase 3 Clinical Trials. Neurol Ther. 2025 Dec;14(6):2491-2506. doi: 10.1007/s40120-025-00827-6. Epub 2025 Oct 4. PMID 41045349
- [Derived] Chaudhuri KR, Facheris MF, Bergmans B, Bergquist F, Criswell SR, Jia J, Kukreja P, Mukai Y, Spiegel AM, Gupta R, Bergmann L, Pahwa R. Improved Sleep Correlates with Improved Quality of Life and Motor Symptoms with Foslevodopa/Foscarbidopa. Mov Disord Clin Pract. 2024 Jul;11(7):861-866. doi: 10.1002/mdc3.14018. Epub 2024 Mar 11. PMID 38465885
- [Derived] Aldred J, Freire-Alvarez E, Amelin AV, Antonini A, Bergmans B, Bergquist F, Bouchard M, Budur K, Carroll C, Chaudhuri KR, Criswell SR, Danielsen EH, Gandor F, Jia J, Kimber TE, Mochizuki H, Robieson WZ, Spiegel AM, Standaert DG, Talapala S, Facheris MF, Fung VSC. Continuous Subcutaneous Foslevodopa/Foscarbidopa in Parkinson's Disease: Safety and Efficacy Results From a 12-Month, Single-Arm, Open-Label, Phase 3 Study. Neurol Ther. 2023 Dec;12(6):1937-1958. doi: 10.1007/s40120-023-00533-1. Epub 2023 Aug 26. PMID 37632656

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All enrolled participants
Period: Overall Study
Arm/Group | ABBV-951 Low Dose Subgroup | ABBV-951 High Dose Subgroup
Started | 131 | 113
Completed | 84 | 65
Not Completed | 47 | 48
Not completed — Adverse Event | 23 | 25
Not completed — Withdrew consent | 16 | 12
Not completed — Lost to Follow-up | 0 | 1
Not completed — Lack of Efficacy | 4 | 5
Not completed — Difficulty with drug delivery system | 2 | 3
Not completed — Other, not specified | 2 | 2

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set: all participants who received any ABBV-951 infusion
Groups:
- Total: Total of all reporting groups
Arm/Group | ABBV-951 Low Dose Subgroup | ABBV-951 High Dose Subgroup | Total
Number analyzed (Participants) | 131 | 113 | 244
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.5 (8.87) | 64.4 (9.54) | 63.9 (9.18)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 66 | 32 | 98
  Male | 65 | 81 | 146
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 12 | 20
  Not Hispanic or Latino | 123 | 101 | 224
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 27 | 7 | 34
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 102 | 105 | 207
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events
Description: An adverse event (AE) is defined as any untoward medical occurrence in a patient or clinical investigation participant administered a pharmaceutical product which does not necessarily have a causal relationship with this treatment. The investigator assesses the relationship of each event to the use of study drug. A serious adverse event (SAE) is an event that results in death, is life-threatening, requires or prolongs hospitalization, results in a congenital anomaly, persistent or significant disability/incapacity or is an important medical event that, based on medical judgment, may jeopardize the participant and may require medical or surgical intervention to prevent any of the outcomes listed above. Treatment-emergent adverse events/treatment-emergent serious adverse events (TEAEs/TESAEs) are defined as any event that began or worsened in severity on or after the first dose of study drug.
Time Frame: From first dose of study drug until 30 days following last dose of study drug (up to 480 days)
Population: Safety Analysis Set: all participants who received any ABBV-951 infusion
Measure: Count of Participants; unit: Participants
Groups:
- ABBV-951 All Participants: After a 4-week Optimization Period, participants continued receiving ABBV-951 by continuous subcutaneous infusion (CSCI) during the 48-week Maintenance Period.
Arm/Group | ABBV-951 Low Dose Subgroup | ABBV-951 High Dose Subgroup | ABBV-951 All Participants
Number analyzed (Participants) | 131 | 113 | 244
Participants
  Any TEAE | 121 | 109 | 230
  TESAE | 32 | 31 | 63

2. Primary Outcome: Number of Participants With Adverse Events of Special Interest
Description: Treatment emergent adverse events of special interest are defined as any adverse event of infusion site infections, infusion site reactions, hallucinations/psychosis, falls and associated injuries, polyneuropathy (peripheral neuropathy), weight loss, or somnolence from the first dose of study drug until 30 days following last dose of study drug.
Time Frame: From first dose of study drug until 30 days following last dose of study drug (up to 480 days)
Population: Safety Analysis Set: all participants who received any ABBV-951 infusion
Measure: Count of Participants; unit: Participants
Arm/Group | ABBV-951 Low Dose Subgroup | ABBV-951 High Dose Subgroup | ABBV-951 All Participants
Number analyzed (Participants) | 131 | 113 | 244
Participants
  Infusion site infections | 42 | 44 | 86
  Infusion site reactions | 103 | 97 | 200
  Hallucinations/psychosis | 32 | 29 | 61
  Falls and associated injuries | 37 | 37 | 74
  Polyneuropathy (peripheral neuropathy) | 14 | 13 | 27
  Weight loss | 12 | 15 | 27
  Somnolence | 9 | 3 | 12

3. Primary Outcome: Number of Participants With Numeric Grade Equal to or Higher Than 5 and With Letter Grade Equal to or Higher Than D on the Infusion Site Evaluation Scale
Description: Skin tolerability was assessed using the Infusion Site Evaluation Scale, a 2-part numeric (0-7) and letter (A-G) grade scale, where a notable skin reaction is defined as a reaction with a numeric grade of 6 or 7 or a letter grade of D, E, F, or G. Any observation of infusion site reaction with irritation criteria > 2 or > C was recorded as an adverse event (AE).
Time Frame: Day 1, Day 2, Week 1, Week 2, Week 3, Week 4, Week 6, Week 13, Week 26, Week 39, and Week 52
Population: Safety Analysis Set: all participants who received any ABBV-951 infusion
Measure: Count of Participants; unit: Participants
Arm/Group | ABBV-951 Low Dose Subgroup | ABBV-951 High Dose Subgroup | ABBV-951 All Participants
Number analyzed (Participants) | 131 | 113 | 244
Participants | 10 | 15 | 25

4. Primary Outcome: Hematocrit (Hematology): Change From Baseline to End of Study
Description: Samples for clinical laboratory tests were collected at study visits, and a certified central laboratory was used to process the samples and provide results.
Time Frame: Baseline, Weeks 6, 26, 39, and 52
Population: Safety Analysis Set: all participants who received any ABBV-951 infusion with available data
Measure: Mean (Standard Deviation); unit: proportion of red blood cells in blood
Arm/Group | ABBV-951 Low Dose Subgroup | ABBV-951 High Dose Subgroup | ABBV-951 All Participants
Number analyzed (Participants) | 128 | 113 | 241
proportion of red blood cells in blood
  Week 6: number analyzed (Participants) | 94 | 91 | 185
  Week 6 | -0.02 (0.031) | -0.02 (0.029) | -0.02 (0.030)
  Week 26: number analyzed (Participants) | 69 | 61 | 130
  Week 26 | -0.01 (0.030) | -0.02 (0.026) | -0.02 (0.028)
  Week 39: number analyzed (Participants) | 61 | 53 | 114
  Week 39 | -0.02 (0.028) | -0.02 (0.029) | -0.02 (0.028)
  Week 52: number analyzed (Participants) | 62 | 56 | 118
  Week 52 | -0.02 (0.029) | -0.02 (0.028) | -0.02 (0.029)

5. Primary Outcome: Hemoglobin (Hematology): Change From Baseline to End of Study
Description: as for outcome 4
Time Frame: Baseline, Weeks 6, 26, 39, and 52
Population: Safety Analysis Set: all participants who received any ABBV-951 infusion with available data
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | ABBV-951 Low Dose Subgroup | ABBV-951 High Dose Subgroup | ABBV-951 All Participants
Number analyzed (Participants) | 130 | 113 | 243
g/L
  Week 6: number analyzed (Participants) | 98 | 93 | 191
  Week 6 | -5.00 (8.308) | -6.82 (9.222) | -5.89 (8.789)
  Week 26: number analyzed (Participants) | 71 | 63 | 134
  Week 26 | -5.42 (9.296) | -4.48 (7.502) | -4.98 (8.482)
  Week 39: number analyzed (Participants) | 68 | 53 | 121
  Week 39 | -5.74 (8.430) | -6.58 (8.601) | -6.11 (8.480)
  Week 52: number analyzed (Participants) | 69 | 56 | 125
  Week 52 | -7.96 (8.862) | -5.80 (9.308) | -6.99 (9.091)

6. Primary Outcome: Red Blood Cell (RBC) Count (Hematology): Change From Baseline to End of Study
Description: as for outcome 4
Time Frame: Baseline, Weeks 6, 26, 39, and 52
Population: Safety Analysis Set: all participants who received any ABBV-951 infusion with available data
Measure: Mean (Standard Deviation); unit: cells*10^12/L
Arm/Group | ABBV-951 Low Dose Subgroup | ABBV-951 High Dose Subgroup | ABBV-951 All Participants
Number analyzed (Participants) | 130 | 113 | 243
cells*10^12/L
  Week 6: number analyzed (Participants) | 96 | 93 | 189
  Week 6 | -0.15 (0.261) | -0.21 (0.296) | -0.18 (0.280)
  Week 26: number analyzed (Participants) | 71 | 63 | 134
  Week 26 | -0.12 (0.295) | -0.13 (0.273) | -0.13 (0.284)
  Week 39: number analyzed (Participants) | 68 | 53 | 121
  Week 39 | -0.14 (0.271) | -0.19 (0.290) | -0.17 (0.279)
  Week 52: number analyzed (Participants) | 69 | 56 | 125
  Week 52 | -0.21 (0.291) | -0.16 (0.293) | -0.19 (0.292)

7. Primary Outcome: White Blood Cell (WBC) Count (Hematology): Change From Baseline to End of Study
Description: as for outcome 4
Time Frame: Baseline, Weeks 6, 26, 39, and 52
Population: Safety Analysis Set: all participants who received any ABBV-951 infusion with available data
Measure: Mean (Standard Deviation); unit: cells*10^9/L
Arm/Group | ABBV-951 Low Dose Subgroup | ABBV-951 High Dose Subgroup | ABBV-951 All Participants
Number analyzed (Participants) | 130 | 113 | 243
cells*10^9/L
  Week 6: number analyzed (Participants) | 98 | 93 | 191
  Week 6 | 0.02 (1.705) | 0.32 (2.120) | 0.17 (1.919)
  Week 26: number analyzed (Participants) | 71 | 63 | 134
  Week 26 | 0.12 (1.892) | 0.22 (2.990) | 0.17 (2.460)
  Week 39: number analyzed (Participants) | 69 | 53 | 122
  Week 39 | 0.35 (4.014) | 0.38 (1.670) | 0.36 (3.202)
  Week 52: number analyzed (Participants) | 69 | 56 | 125
  Week 52 | -0.08 (2.027) | -0.04 (1.568) | -0.06 (1.829)

8. Primary Outcome: Neutrophils (Hematology): Change From Baseline to End of Study
Description: as for outcome 4
Time Frame: Baseline, Weeks 6, 26, 39, and 52
Population: Safety Analysis Set: all participants who received any ABBV-951 infusion with available data
Measure: Mean (Standard Deviation); unit: cells*10^9/L
Arm/Group | ABBV-951 Low Dose Subgroup | ABBV-951 High Dose Subgroup | ABBV-951 All Participants
Number analyzed (Participants) | 130 | 113 | 243
cells*10^9/L
  Week 6: number analyzed (Participants) | 97 | 92 | 189
  Week 6 | 0.01 (1.720) | 0.33 (2.102) | 0.17 (1.917)
  Week 26: number analyzed (Participants) | 71 | 63 | 134
  Week 26 | -0.03 (1.813) | 143.08 (1133.988) | 67.25 (777.558)
  Week 39: number analyzed (Participants) | 68 | 53 | 121
  Week 39 | -0.23 (2.380) | 0.18 (1.635) | -0.05 (2.089)
  Week 52: number analyzed (Participants) | 69 | 56 | 125
  Week 52 | -0.14 (1.986) | -0.04 (1.498) | -0.10 (1.778)

9. Primary Outcome: Lymphocytes (Hematology): Change From Baseline to End of Study
Description: as for outcome 4
Time Frame: Baseline, Weeks 6, 26, 39, and 52
Population: Safety Analysis Set: all participants who received any ABBV-951 infusion with available data
Measure: Mean (Standard Deviation); unit: cells*10^9/L
Arm/Group | ABBV-951 Low Dose Subgroup | ABBV-951 High Dose Subgroup | ABBV-951 All Participants
Number analyzed (Participants) | 130 | 113 | 243
cells*10^9/L
  Week 6: number analyzed (Participants) | 97 | 92 | 189
  Week 6 | 0.06 (0.305) | -0.07 (0.326) | 0.00 (0.321)
  Week 26: number analyzed (Participants) | 71 | 63 | 134
  Week 26 | 0.09 (0.331) | 13.92 (110.588) | 6.59 (75.823)
  Week 39: number analyzed (Participants) | 68 | 53 | 121
  Week 39 | 0.03 (0.394) | 0.04 (0.312) | 0.03 (0.359)
  Week 52: number analyzed (Participants) | 69 | 56 | 125
  Week 52 | 0.04 (0.394) | -0.05 (0.294) | 0.00 (0.354)

10. Primary Outcome: Monocytes (Hematology): Change From Baseline to End of Study
Description: as for outcome 4
Time Frame: Baseline, Weeks 6, 26, 39, and 52
Population: Safety Analysis Set: all participants who received any ABBV-951 infusion with available data
Measure: Mean (Standard Deviation); unit: cells*10^9/L
Arm/Group | ABBV-951 Low Dose Subgroup | ABBV-951 High Dose Subgroup | ABBV-951 All Participants
Number analyzed (Participants) | 130 | 113 | 243
cells*10^9/L
  Week 6: number analyzed (Participants) | 96 | 92 | 188
  Week 6 | 0.01 (0.127) | 0.01 (0.123) | 0.01 (0.125)
  Week 26: number analyzed (Participants) | 71 | 63 | 134
  Week 26 | 0.02 (0.095) | 17.43 (138.498) | 8.21 (94.963)
  Week 39: number analyzed (Participants) | 68 | 53 | 121
  Week 39 | 0.02 (0.120) | 0.03 (0.122) | 0.02 (0.120)
  Week 52: number analyzed (Participants) | 69 | 56 | 125
  Week 52 | 0.00 (0.109) | 0.01 (0.132) | 0.00 (0.119)

11. Primary Outcome: Absolute Platelet Count (Hematology): Change From Baseline to End of Study
Description: as for outcome 4
Time Frame: Baseline, Weeks 6, 26, 39, and 52
Population: Safety Analysis Set: all participants who received any ABBV-951 infusion with available data
Measure: Mean (Standard Deviation); unit: cells*10^9/L
Arm/Group | ABBV-951 Low Dose Subgroup | ABBV-951 High Dose Subgroup | ABBV-951 All Participants
Number analyzed (Participants) | 130 | 112 | 242
cells*10^9/L
  Week 6: number analyzed (Participants) | 96 | 92 | 188
  Week 6 | 4.59 (36.489) | 0.39 (40.844) | 2.54 (38.635)
  Week 26: number analyzed (Participants) | 71 | 62 | 133
  Week 26 | -1.68 (43.279) | -10.39 (43.757) | -5.74 (43.556)
  Week 39: number analyzed (Participants) | 68 | 52 | 120
  Week 39 | -3.90 (43.848) | -7.29 (49.222) | -5.37 (46.084)
  Week 52: number analyzed (Participants) | 69 | 54 | 123
  Week 52 | -3.41 (41.120) | -10.63 (44.537) | -6.58 (42.628)

12. Primary Outcome: Mean Corpuscular Hemoglobin (Hematology): Change From Baseline to End of Study
Description: as for outcome 4
Time Frame: Baseline, Weeks 6, 26, 39, and 52
Population: Safety Analysis Set: all participants who received any ABBV-951 infusion with available data
Measure: Mean (Standard Deviation); unit: picograms
Arm/Group | ABBV-951 Low Dose Subgroup | ABBV-951 High Dose Subgroup | ABBV-951 All Participants
Number analyzed (Participants) | 130 | 113 | 243
picograms
  Week 6: number analyzed (Participants) | 96 | 92 | 188
  Week 6 | -0.09 (0.822) | -0.15 (0.825) | -0.12 (0.821)
  Week 26: number analyzed (Participants) | 71 | 62 | 133
  Week 26 | -0.38 (1.033) | 0.05 (1.078) | -0.18 (1.072)
  Week 39: number analyzed (Participants) | 68 | 53 | 121
  Week 39 | -0.34 (1.205) | -0.08 (0.978) | -0.22 (1.114)
  Week 52: number analyzed (Participants) | 69 | 56 | 125
  Week 52 | -0.36 (1.124) | -0.07 (1.142) | -0.23 (1.137)

13. Primary Outcome: Mean Corpuscular Volume Concentration (MCHC) (Hematology): Change From Baseline to End of Study
Description: as for outcome 4
Time Frame: Baseline, Weeks 6, 26, 39, and 52
Population: Safety Analysis Set: all participants who received any ABBV-951 infusion with available data
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | ABBV-951 Low Dose Subgroup | ABBV-951 High Dose Subgroup | ABBV-951 All Participants
Number analyzed (Participants) | 128 | 113 | 241
g/L
  Week 6: number analyzed (Participants) | 93 | 90 | 183
  Week 6 | 2.15 (11.689) | 1.78 (10.870) | 1.97 (11.264)
  Week 26: number analyzed (Participants) | 69 | 60 | 129
  Week 26 | -1.30 (14.844) | 2.17 (15.741) | 0.31 (15.306)
  Week 39: number analyzed (Participants) | 61 | 53 | 114
  Week 39 | -2.13 (13.677) | -2.64 (14.826) | -2.37 (14.161)
  Week 52: number analyzed (Participants) | 62 | 56 | 118
  Week 52 | -0.16 (12.609) | 0.18 (13.684) | 0.00 (13.074)

14. Primary Outcome: Prothrombin Time (PT) (Hematology): Change From Baseline to End of Study
Description: as for outcome 4
Time Frame: Baseline, Weeks 6, 26, 39, and 52
Population: Safety Analysis Set: all participants who received any ABBV-951 infusion with available data
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | ABBV-951 Low Dose Subgroup | ABBV-951 High Dose Subgroup | ABBV-951 All Participants
Number analyzed (Participants) | 131 | 113 | 244
seconds
  Week 6: number analyzed (Participants) | 100 | 93 | 193
  Week 6 | 0.03 (0.480) | -0.09 (2.556) | -0.03 (1.803)
  Week 26: number analyzed (Participants) | 70 | 57 | 127
  Week 26 | -0.08 (1.026) | -0.36 (3.187) | -0.20 (2.261)
  Week 39: number analyzed (Participants) | 70 | 51 | 121
  Week 39 | 0.10 (0.569) | -0.21 (3.396) | -0.03 (2.239)
  Week 52: number analyzed (Participants) | 72 | 52 | 124
  Week 52 | 0.10 (0.889) | -0.22 (3.703) | -0.04 (2.483)

15. Primary Outcome: Activated Partial Thromboplastin Time (Hematology): Change From Baseline to End of Study
Description: as for outcome 4
Time Frame: Baseline, Weeks 6, 26, 39, and 52
Population: Safety Analysis Set: all participants who received any ABBV-951 infusion with available data
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | ABBV-951 Low Dose Subgroup | ABBV-951 High Dose Subgroup | ABBV-951 All Participants
Number analyzed (Participants) | 131 | 113 | 244
seconds
  Week 6: number analyzed (Participants) | 100 | 93 | 193
  Week 6 | -0.27 (2.151) | 0.55 (2.483) | 0.13 (2.347)
  Week 26: number analyzed (Participants) | 70 | 57 | 127
  Week 26 | -0.02 (1.898) | 0.48 (1.932) | 0.20 (1.922)
  Week 39: number analyzed (Participants) | 70 | 51 | 121
  Week 39 | 0.14 (1.556) | 0.67 (3.672) | 0.36 (2.661)
  Week 52: number analyzed (Participants) | 71 | 51 | 122
  Week 52 | -0.09 (2.156) | 0.88 (2.992) | 0.32 (2.573)

16. Primary Outcome: Blood Urea Nitrogen (BUN) (Clinical Chemistry): Change From Baseline to End of Study
Description: as for outcome 4
Time Frame: Baseline, Weeks 6, 26, 39, and 52
Population: Safety Analysis Set: all participants who received any ABBV-951 infusion with available data
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | ABBV-951 Low Dose Subgroup | ABBV-951 High Dose Subgroup | ABBV-951 All Participants
Number analyzed (Participants) | 131 | 113 | 244
mmol/L
  Week 6: number analyzed (Participants) | 103 | 96 | 199
  Week 6 | 0.02 (1.348) | -0.01 (1.560) | 0.00 (1.450)
  Week 26: number analyzed (Participants) | 75 | 62 | 137
  Week 26 | 0.21 (1.489) | 0.17 (1.600) | 0.19 (1.535)
  Week 39: number analyzed (Participants) | 72 | 55 | 127
  Week 39 | 0.41 (1.852) | 0.05 (1.659) | 0.25 (1.773)
  Week 52: number analyzed (Participants) | 74 | 56 | 130
  Week 52 | 0.16 (1.836) | 0.15 (1.342) | 0.16 (1.636)

17. Primary Outcome: Creatinine (Clinical Chemistry): Change From Baseline to End of Study
Description: as for outcome 4
Time Frame: Baseline, Weeks 6, 26, 39, and 52
Population: Safety Analysis Set: all participants who received any ABBV-951 infusion with available data
Measure: Mean (Standard Deviation); unit: µmol/L
Arm/Group | ABBV-951 Low Dose Subgroup | ABBV-951 High Dose Subgroup | ABBV-951 All Participants
Number analyzed (Participants) | 131 | 113 | 244
µmol/L
  Week 6: number analyzed (Participants) | 104 | 96 | 200
  Week 6 | -4.45 (9.227) | -5.67 (10.725) | -5.04 (9.968)
  Week 26: number analyzed (Participants) | 75 | 63 | 138
  Week 26 | -2.71 (10.478) | -4.07 (12.074) | -3.33 (11.213)
  Week 39: number analyzed (Participants) | 72 | 55 | 127
  Week 39 | -1.47 (12.414) | -4.02 (10.182) | -2.58 (11.527)
  Week 52: number analyzed (Participants) | 74 | 56 | 130
  Week 52 | -4.78 (11.446) | -5.21 (9.941) | -4.96 (10.785)

18. Primary Outcome: Creatine Phosphokinase (Clinical Chemistry): Change From Baseline to End of Study
Description: as for outcome 4
Time Frame: Baseline, Weeks 6, 26, 39, and 52
Population: Safety Analysis Set: all participants who received any ABBV-951 infusion with available data
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | ABBV-951 Low Dose Subgroup | ABBV-951 High Dose Subgroup | ABBV-951 All Participants
Number analyzed (Participants) | 131 | 113 | 244
U/L
  Week 6: number analyzed (Participants) | 103 | 96 | 199
  Week 6 | 2.52 (56.209) | -11.01 (94.662) | -4.01 (77.285)
  Week 26: number analyzed (Participants) | 75 | 61 | 136
  Week 26 | 5.61 (51.627) | -15.44 (62.435) | -3.83 (57.480)
  Week 39: number analyzed (Participants) | 72 | 54 | 126
  Week 39 | 8.40 (96.021) | -9.67 (75.655) | 0.66 (88.002)
  Week 52: number analyzed (Participants) | 74 | 56 | 130
  Week 52 | 30.39 (125.044) | -16.55 (85.305) | 10.17 (111.783)

19. Primary Outcome: Total Bilirubin (Clinical Chemistry): Change From Baseline to End of Study
Description: as for outcome 4
Time Frame: Baseline, Weeks 6, 26, 39, and 52
Population: Safety Analysis Set: all participants who received any ABBV-951 infusion with available data
Measure: Mean (Standard Deviation); unit: µmol/L
Arm/Group | ABBV-951 Low Dose Subgroup | ABBV-951 High Dose Subgroup | ABBV-951 All Participants
Number analyzed (Participants) | 131 | 113 | 244
µmol/L
  Week 6: number analyzed (Participants) | 103 | 96 | 199
  Week 6 | -0.85 (3.420) | -0.15 (3.167) | -0.51 (3.311)
  Week 26: number analyzed (Participants) | 75 | 61 | 136
  Week 26 | -0.43 (3.535) | 0.28 (2.814) | -0.11 (3.240)
  Week 39: number analyzed (Participants) | 72 | 55 | 127
  Week 39 | -0.71 (2.881) | 0.31 (3.754) | -0.27 (3.313)
  Week 52: number analyzed (Participants) | 74 | 56 | 130
  Week 52 | -0.30 (3.673) | -0.15 (3.250) | -0.24 (3.485)

20. Primary Outcome: Serum Alanine Aminotransferase (Clinical Chemistry): Change From Baseline to End of Study
Description: as for outcome 4
Time Frame: Baseline, Weeks 6, 26, 39, and 52
Population: Safety Analysis Set: all participants who received any ABBV-951 infusion with available data
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | ABBV-951 Low Dose Subgroup | ABBV-951 High Dose Subgroup | ABBV-951 All Participants
Number analyzed (Participants) | 131 | 113 | 244
U/L
  Week 6: number analyzed (Participants) | 103 | 96 | 199
  Week 6 | -8.94 (8.928) | -11.28 (10.053) | -10.07 (9.535)
  Week 26: number analyzed (Participants) | 75 | 61 | 136
  Week 26 | -8.95 (9.869) | -11.66 (11.294) | -10.16 (10.579)
  Week 39: number analyzed (Participants) | 71 | 54 | 125
  Week 39 | -9.70 (9.145) | -10.09 (13.476) | -9.87 (11.175)
  Week 52: number analyzed (Participants) | 73 | 56 | 129
  Week 52 | -9.37 (10.347) | -12.11 (9.947) | -10.56 (10.227)

21. Primary Outcome: Serum Aspartate Aminotransferase (Clinical Chemistry): Change From Baseline to End of Study
Description: as for outcome 4
Time Frame: Baseline, Weeks 6, 26, 39, and 52
Population: Safety Analysis Set: all participants who received any ABBV-951 infusion with available data
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | ABBV-951 Low Dose Subgroup | ABBV-951 High Dose Subgroup | ABBV-951 All Participants
Number analyzed (Participants) | 131 | 113 | 244
U/L
  Week 6: number analyzed (Participants) | 102 | 95 | 197
  Week 6 | -1.89 (4.881) | -2.21 (6.163) | -2.05 (5.524)
  Week 26: number analyzed (Participants) | 74 | 59 | 133
  Week 26 | -0.69 (8.569) | -2.56 (7.013) | -1.52 (7.943)
  Week 39: number analyzed (Participants) | 72 | 54 | 126
  Week 39 | -1.38 (6.714) | -1.17 (7.036) | -1.29 (6.827)
  Week 52: number analyzed (Participants) | 73 | 55 | 128
  Week 52 | -0.81 (6.576) | -0.82 (7.794) | -0.81 (7.095)

22. Primary Outcome: Serum Lactate Dehydrogenase (LDH) (Clinical Chemistry): Change From Baseline to End of Study
Description: as for outcome 4
Time Frame: Baseline, Weeks 6, 26, 39, and 52
Population: Safety Analysis Set: all participants who received any ABBV-951 infusion with available data
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | ABBV-951 Low Dose Subgroup | ABBV-951 High Dose Subgroup | ABBV-951 All Participants
Number analyzed (Participants) | 129 | 109 | 238
U/L
  Week 6: number analyzed (Participants) | 93 | 89 | 182
  Week 6 | -6.57 (26.734) | -8.58 (23.626) | -7.55 (25.213)
  Week 26: number analyzed (Participants) | 67 | 56 | 123
  Week 26 | -1.66 (23.894) | -4.91 (23.613) | -3.14 (23.725)
  Week 39: number analyzed (Participants) | 59 | 47 | 106
  Week 39 | -2.17 (25.010) | -2.02 (26.431) | -2.10 (25.526)
  Week 52: number analyzed (Participants) | 71 | 47 | 118
  Week 52 | 0.14 (22.788) | 3.32 (26.413) | 1.41 (24.237)

23. Primary Outcome: Gamma-glutamyl Transferase (Clinical Chemistry): Change From Baseline to End of Study
Description: as for outcome 4
Time Frame: Baseline, Weeks 6, 26, 39, and 52
Population: Safety Analysis Set: all participants who received any ABBV-951 infusion with available data
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | ABBV-951 Low Dose Subgroup | ABBV-951 High Dose Subgroup | ABBV-951 All Participants
Number analyzed (Participants) | 131 | 113 | 244
U/L
  Week 6: number analyzed (Participants) | 103 | 96 | 199
  Week 6 | -1.07 (9.516) | -3.13 (9.393) | -2.06 (9.489)
  Week 26: number analyzed (Participants) | 75 | 62 | 137
  Week 26 | -1.47 (11.487) | -5.02 (15.370) | -3.07 (13.450)
  Week 39: number analyzed (Participants) | 72 | 54 | 126
  Week 39 | -1.92 (10.860) | -4.67 (12.516) | -3.10 (11.631)
  Week 52: number analyzed (Participants) | 74 | 56 | 130
  Week 52 | 1.69 (23.235) | -3.09 (14.538) | -0.37 (20.031)

24. Primary Outcome: Alkaline Phosphatase (Clinical Chemistry): Change From Baseline to End of Study
Description: as for outcome 4
Time Frame: Baseline, Weeks 6, 26, 39, and 52
Population: Safety Analysis Set: all participants who received any ABBV-951 infusion with available data
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | ABBV-951 Low Dose Subgroup | ABBV-951 High Dose Subgroup | ABBV-951 All Participants
Number analyzed (Participants) | 131 | 113 | 244
U/L
  Week 6: number analyzed (Participants) | 103 | 96 | 199
  Week 6 | -1.91 (12.394) | -4.56 (12.340) | -3.19 (12.408)
  Week 26: number analyzed (Participants) | 75 | 63 | 138
  Week 26 | 1.68 (18.995) | -2.86 (14.157) | -0.39 (17.051)
  Week 39: number analyzed (Participants) | 72 | 55 | 127
  Week 39 | -2.28 (12.252) | -5.02 (16.088) | -3.46 (14.049)
  Week 52: number analyzed (Participants) | 74 | 56 | 130
  Week 52 | 0.55 (18.637) | -1.54 (13.796) | -0.35 (16.697)

25. Primary Outcome: Sodium (Clinical Chemistry): Change From Baseline to End of Study
Description: as for outcome 4
Time Frame: Baseline, Weeks 6, 26, 39, and 52
Population: Safety Analysis Set: all participants who received any ABBV-951 infusion with available data
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | ABBV-951 Low Dose Subgroup | ABBV-951 High Dose Subgroup | ABBV-951 All Participants
Number analyzed (Participants) | 131 | 113 | 244
mmol/L
  Week 6: number analyzed (Participants) | 103 | 95 | 198
  Week 6 | -0.52 (3.168) | -1.06 (2.592) | -0.78 (2.911)
  Week 26: number analyzed (Participants) | 74 | 61 | 135
  Week 26 | -0.35 (3.173) | -1.26 (2.744) | -0.76 (3.010)
  Week 39: number analyzed (Participants) | 72 | 53 | 125
  Week 39 | -0.90 (2.984) | -0.68 (2.772) | -0.81 (2.887)
  Week 52: number analyzed (Participants) | 73 | 56 | 129
  Week 52 | -0.55 (2.774) | -0.84 (2.164) | -0.67 (2.522)

26. Primary Outcome: Potassium (Clinical Chemistry): Change From Baseline to End of Study
Description: as for outcome 4
Time Frame: Baseline, Weeks 6, 26, 39, and 52
Population: Safety Analysis Set: all participants who received any ABBV-951 infusion with available data
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | ABBV-951 Low Dose Subgroup | ABBV-951 High Dose Subgroup | ABBV-951 All Participants
Number analyzed (Participants) | 131 | 113 | 244
mmol/L
  Week 6: number analyzed (Participants) | 103 | 96 | 199
  Week 6 | -0.02 (0.335) | -0.08 (0.330) | -0.05 (0.333)
  Week 26: number analyzed (Participants) | 74 | 61 | 135
  Week 26 | 0.01 (0.367) | 0.00 (0.373) | 0.00 (0.368)
  Week 39: number analyzed (Participants) | 72 | 52 | 124
  Week 39 | -0.01 (0.389) | -0.09 (0.382) | -0.04 (0.387)
  Week 52: number analyzed (Participants) | 73 | 56 | 129
  Week 52 | -0.10 (0.369) | -0.03 (0.338) | -0.07 (0.357)

27. Primary Outcome: Calcium (Clinical Chemistry): Change From Baseline to End of Study
Description: as for outcome 4
Time Frame: Baseline, Weeks 6, 26, 39, and 52
Population: Safety Analysis Set: all participants who received any ABBV-951 infusion with available data
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | ABBV-951 Low Dose Subgroup | ABBV-951 High Dose Subgroup | ABBV-951 All Participants
Number analyzed (Participants) | 131 | 113 | 244
mmol/L
  Week 6: number analyzed (Participants) | 103 | 96 | 199
  Week 6 | -0.02 (0.079) | -0.04 (0.086) | -0.03 (0.083)
  Week 26: number analyzed (Participants) | 75 | 63 | 138
  Week 26 | -0.03 (0.080) | -0.04 (0.091) | -0.03 (0.085)
  Week 39: number analyzed (Participants) | 72 | 55 | 127
  Week 39 | -0.04 (0.091) | -0.05 (0.087) | -0.05 (0.089)
  Week 52: number analyzed (Participants) | 74 | 56 | 130
  Week 52 | -0.06 (0.084) | -0.04 (0.092) | -0.05 (0.088)

28. Primary Outcome: Inorganic Phosphorus (Clinical Chemistry): Change From Baseline to End of Study
Description: as for outcome 4
Time Frame: Baseline, Weeks 6, 26, 39, and 52
Population: Safety Analysis Set: all participants who received any ABBV-951 infusion with available data
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | ABBV-951 Low Dose Subgroup | ABBV-951 High Dose Subgroup | ABBV-951 All Participants
Number analyzed (Participants) | 131 | 113 | 244
mmol/L
  Week 6: number analyzed (Participants) | 103 | 96 | 199
  Week 6 | 0.08 (0.173) | 0.08 (0.168) | 0.08 (0.170)
  Week 26: number analyzed (Participants) | 75 | 62 | 137
  Week 26 | 0.09 (0.182) | 0.09 (0.170) | 0.09 (0.176)
  Week 39: number analyzed (Participants) | 72 | 55 | 127
  Week 39 | 0.07 (0.165) | 0.08 (0.155) | 0.08 (0.160)
  Week 52: number analyzed (Participants) | 74 | 56 | 130
  Week 52 | 0.09 (0.169) | 0.08 (0.172) | 0.08 (0.170)

29. Primary Outcome: Uric Acid (Clinical Chemistry): Change From Baseline to End of Study
Description: as for outcome 4
Time Frame: Baseline, Weeks 6, 26, 39, and 52
Population: Safety Analysis Set: all participants who received any ABBV-951 infusion with available data
Measure: Mean (Standard Deviation); unit: µmol/L
Arm/Group | ABBV-951 Low Dose Subgroup | ABBV-951 High Dose Subgroup | ABBV-951 All Participants
Number analyzed (Participants) | 131 | 113 | 244
µmol/L
  Week 6: number analyzed (Participants) | 103 | 96 | 199
  Week 6 | -28.36 (51.219) | -37.43 (37.302) | -32.73 (45.163)
  Week 26: number analyzed (Participants) | 75 | 62 | 137
  Week 26 | -16.66 (60.922) | -32.91 (34.446) | -24.01 (51.163)
  Week 39: number analyzed (Participants) | 72 | 55 | 127
  Week 39 | -13.55 (57.830) | -35.80 (40.965) | -23.18 (52.213)
  Week 52: number analyzed (Participants) | 74 | 56 | 130
  Week 52 | -15.27 (56.459) | -31.23 (29.780) | -22.15 (47.380)

30. Primary Outcome: Total Cholesterol (Clinical Chemistry): Change From Baseline to End of Study
Description: as for outcome 4
Time Frame: Baseline, Weeks 6, 26, 39, and 52
Population: Safety Analysis Set: all participants who received any ABBV-951 infusion with available data
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | ABBV-951 Low Dose Subgroup | ABBV-951 High Dose Subgroup | ABBV-951 All Participants
Number analyzed (Participants) | 131 | 113 | 244
mmol/L
  Week 6: number analyzed (Participants) | 102 | 95 | 197
  Week 6 | -0.37 (0.688) | -0.57 (0.556) | -0.47 (0.634)
  Week 26: number analyzed (Participants) | 74 | 62 | 136
  Week 26 | -0.19 (0.657) | -0.31 (0.661) | -0.25 (0.659)
  Week 39: number analyzed (Participants) | 72 | 53 | 125
  Week 39 | -0.33 (0.565) | -0.41 (0.552) | -0.36 (0.559)
  Week 52: number analyzed (Participants) | 73 | 56 | 129
  Week 52 | -0.31 (0.660) | -0.25 (0.594) | -0.29 (0.630)

31. Primary Outcome: Albumin (Clinical Chemistry): Change From Baseline to End of Study
Description: as for outcome 4
Time Frame: Baseline, Weeks 6, 26, 39, and 52
Population: Safety Analysis Set: all participants who received any ABBV-951 infusion with available data
Measure: Mean (Standard Deviation); unit: g/L
Arm/Group | ABBV-951 Low Dose Subgroup | ABBV-951 High Dose Subgroup | ABBV-951 All Participants
Number analyzed (Participants) | 131 | 113 | 244
g/L
  Week 6: number analyzed (Participants) | 103 | 96 | 199
  Week 6 | -1.65 (2.782) | -1.95 (2.885) | -1.79 (2.829)
  Week 26: number analyzed (Participants) | 75 | 63 | 138
  Week 26 | -1.31 (2.541) | -1.14 (2.558) | -1.23 (2.541)
  Week 39: number analyzed (Participants) | 72 | 55 | 127
  Week 39 | -1.75 (2.782) | -1.56 (2.507) | -1.67 (2.658)
  Week 52: number analyzed (Participants) | 74 | 56 | 130
  Week 52 | -1.96 (2.949) | -1.02 (3.205) | -1.55 (3.086)

32. Primary Outcome: Glucose (Clinical Chemistry): Change From Baseline to End of Study
Description: as for outcome 4
Time Frame: Baseline, Weeks 6, 26, 39, and 52
Population: Safety Analysis Set: all participants who received any ABBV-951 infusion with available data
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | ABBV-951 Low Dose Subgroup | ABBV-951 High Dose Subgroup | ABBV-951 All Participants
Number analyzed (Participants) | 131 | 113 | 244
mmol/L
  Week 6: number analyzed (Participants) | 103 | 97 | 200
  Week 6 | -0.39 (1.186) | -0.39 (1.438) | -0.39 (1.311)
  Week 26: number analyzed (Participants) | 75 | 63 | 138
  Week 26 | -0.37 (1.271) | -0.14 (1.486) | -0.27 (1.373)
  Week 39: number analyzed (Participants) | 72 | 55 | 127
  Week 39 | -0.33 (1.181) | -0.60 (1.327) | -0.45 (1.249)
  Week 52: number analyzed (Participants) | 74 | 56 | 130
  Week 52 | -0.32 (1.917) | -0.55 (1.479) | -0.42 (1.740)

33. Primary Outcome: Sodium Bicarbonate/CO2 (Clinical Chemistry): Change From Baseline to End of Study
Description: as for outcome 4
Time Frame: Baseline, Weeks 6, 26, 39, and 52
Population: Safety Analysis Set: all participants who received any ABBV-951 infusion with available data
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | ABBV-951 Low Dose Subgroup | ABBV-951 High Dose Subgroup | ABBV-951 All Participants
Number analyzed (Participants) | 130 | 113 | 243
mmol/L
  Week 6: number analyzed (Participants) | 100 | 94 | 194
  Week 6 | 1.19 (2.372) | 0.97 (2.518) | 1.09 (2.440)
  Week 26: number analyzed (Participants) | 71 | 60 | 131
  Week 26 | 0.77 (2.418) | 0.28 (2.744) | 0.55 (2.574)
  Week 39: number analyzed (Participants) | 67 | 50 | 117
  Week 39 | 0.90 (2.240) | 0.63 (2.874) | 0.78 (2.522)
  Week 52: number analyzed (Participants) | 72 | 55 | 127
  Week 52 | 0.78 (2.374) | 0.57 (2.304) | 0.69 (2.337)

34. Primary Outcome: Magnesium (Clinical Chemistry): Change From Baseline to End of Study
Description: as for outcome 4
Time Frame: Baseline, Weeks 6, 26, 39, and 52
Population: Safety Analysis Set: all participants who received any ABBV-951 infusion with available data
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | ABBV-951 Low Dose Subgroup | ABBV-951 High Dose Subgroup | ABBV-951 All Participants
Number analyzed (Participants) | 131 | 113 | 244
mmol/L
  Week 6: number analyzed (Participants) | 103 | 95 | 198
  Week 6 | -0.03 (0.067) | -0.03 (0.058) | -0.03 (0.063)
  Week 26: number analyzed (Participants) | 74 | 61 | 135
  Week 26 | -0.03 (0.064) | -0.02 (0.062) | -0.02 (0.063)
  Week 39: number analyzed (Participants) | 72 | 53 | 125
  Week 39 | -0.02 (0.076) | -0.01 (0.073) | -0.02 (0.075)
  Week 52: number analyzed (Participants) | 73 | 56 | 129
  Week 52 | -0.03 (0.078) | -0.01 (0.057) | -0.02 (0.070)

35. Primary Outcome: Creatinine Clearance (Clinical Chemistry): Change From Baseline to End of Study
Description: as for outcome 4
Time Frame: Baseline, Weeks 6, 26, 39, and 52
Population: Safety Analysis Set: all participants who received any ABBV-951 infusion with available data
Measure: Mean (Standard Deviation); unit: mL/sec/1.73m^2
Arm/Group | ABBV-951 Low Dose Subgroup | ABBV-951 High Dose Subgroup | ABBV-951 All Participants
Number analyzed (Participants) | 1 | 1 | 2
mL/sec/1.73m^2
  Week 6 | -0.08 | 0.00 | -0.04 (0.059)
  Week 26: number analyzed (Participants) | 0 | 1 | 1
  Week 26 |  | -0.17 | -0.17
  Week 39: number analyzed (Participants) | 0 | 0 | 0
  Week 52: number analyzed (Participants) | 0 | 0 | 0

36. Primary Outcome: Homocysteine (Clinical Chemistry): Change From Baseline to End of Study
Description: as for outcome 4
Time Frame: Baseline, Weeks 6, 26, and 52
Population: Safety Analysis Set: all participants who received any ABBV-951 infusion with available data
Measure: Mean (Standard Deviation); unit: µmol/L
Arm/Group | ABBV-951 Low Dose Subgroup | ABBV-951 High Dose Subgroup | ABBV-951 All Participants
Number analyzed (Participants) | 131 | 113 | 244
µmol/L
  Week 6: number analyzed (Participants) | 105 | 95 | 200
  Week 6 | 3.07 (5.301) | 6.70 (11.040) | 4.79 (8.692)
  Week 26: number analyzed (Participants) | 76 | 61 | 137
  Week 26 | 4.22 (7.549) | 6.69 (6.306) | 5.32 (7.106)
  Week 52: number analyzed (Participants) | 73 | 52 | 125
  Week 52 | 4.88 (6.103) | 7.24 (8.687) | 5.86 (7.351)

37. Primary Outcome: Vitamin B6 (Clinical Chemistry): Change From Baseline to End of Study
Description: as for outcome 4
Time Frame: Baseline, Weeks 6, 26, and 52
Population: Safety Analysis Set: all participants who received any ABBV-951 infusion with available data
Measure: Mean (Standard Deviation); unit: nmol/L
Arm/Group | ABBV-951 Low Dose Subgroup | ABBV-951 High Dose Subgroup | ABBV-951 All Participants
Number analyzed (Participants) | 131 | 113 | 244
nmol/L
  Week 6: number analyzed (Participants) | 104 | 94 | 198
  Week 6 | 0.30 (129.306) | 4.68 (87.199) | 2.38 (111.069)
  Week 26: number analyzed (Participants) | 76 | 62 | 138
  Week 26 | -4.50 (89.013) | 14.10 (103.462) | 3.86 (95.865)
  Week 52: number analyzed (Participants) | 71 | 54 | 125
  Week 52 | -0.32 (124.059) | 44.30 (124.456) | 18.95 (125.703)

38. Primary Outcome: Vitamin B12 (Clinical Chemistry): Change From Baseline to End of Study
Description: as for outcome 4
Time Frame: Baseline, Weeks 6, 26, and 52
Population: Safety Analysis Set: all participants who received any ABBV-951 infusion with available data
Measure: Mean (Standard Deviation); unit: pmol/L
Groups:
- -ABBV-951 High Dose Subgroup: After a 4-week Optimization Period, participants continued receiving ABBV-951 by continuous subcutaneous infusion (CSCI) during the 48-week Maintenance Period. Participants whose modal total daily dose (most frequent dose) over the entire study was ≥ 2530 mg of Foslevodopa/day were analyzed as the High Dose Subgroup.
Arm/Group | ABBV-951 Low Dose Subgroup | -ABBV-951 High Dose Subgroup | ABBV-951 All Participants
Number analyzed (Participants) | 131 | 113 | 244
pmol/L
  Week 6: number analyzed (Participants) | 104 | 94 | 198
  Week 6 | -229.58 (1349.008) | -206.30 (2217.016) | -218.53 (1808.859)
  Week 26: number analyzed (Participants) | 76 | 63 | 139
  Week 26 | -147.38 (845.662) | -143.30 (1033.488) | -145.53 (931.955)
  Week 52: number analyzed (Participants) | 74 | 54 | 128
  Week 52 | -268.44 (1684.785) | -212.84 (1096.656) | -244.98 (1460.902)

39. Primary Outcome: pH (Urinalysis): Change From Baseline to End of Study
Description: as for outcome 4
Time Frame: Baseline, Weeks 6, 26, 39, and 52
Population: Safety Analysis Set: all participants who received any ABBV-951 infusion with available data
Measure: Mean (Standard Deviation); unit: no units
Arm/Group | ABBV-951 Low Dose Subgroup | ABBV-951 High Dose Subgroup | ABBV-951 All Participants
Number analyzed (Participants) | 131 | 113 | 244
no units
  Week 6: number analyzed (Participants) | 98 | 88 | 186
  Week 6 | 0.07 (0.601) | 0.19 (0.575) | 0.13 (0.590)
  Week 26: number analyzed (Participants) | 69 | 61 | 130
  Week 26 | 0.20 (0.537) | 0.24 (0.560) | 0.22 (0.546)
  Week 39: number analyzed (Participants) | 67 | 54 | 121
  Week 39 | 0.13 (0.566) | 0.31 (0.617) | 0.21 (0.594)
  Week 52: number analyzed (Participants) | 71 | 56 | 127
  Week 52 | 0.18 (0.682) | 0.20 (0.537) | 0.19 (0.620)

40. Primary Outcome: Specific Gravity (Urinalysis): Change From Baseline to End of Study
Description: as for outcome 4
Time Frame: Baseline, Weeks 6, 26, 39, and 52
Population: Safety Analysis Set: all participants who received any ABBV-951 infusion with available data
Measure: Mean (Standard Deviation); unit: No units
Arm/Group | ABBV-951 Low Dose Subgroup | ABBV-951 High Dose Subgroup | ABBV-951 All Participants
Number analyzed (Participants) | 131 | 113 | 244
No units
  Week 6: number analyzed (Participants) | 98 | 88 | 186
  Week 6 | 0.00 (0.009) | 0.00 (0.007) | 0.00 (0.008)
  Week 26: number analyzed (Participants) | 69 | 61 | 130
  Week 26 | 0.00 (0.009) | 0.00 (0.009) | 0.00 (0.009)
  Week 39: number analyzed (Participants) | 68 | 54 | 122
  Week 39 | 0.00 (0.009) | 0.00 (0.009) | 0.00 (0.009)
  Week 52: number analyzed (Participants) | 71 | 56 | 127
  Week 52 | 0.00 (0.010) | 0.00 (0.009) | 0.00 (0.009)

41. Primary Outcome: Orthostatic Systolic Blood Pressure (Vital Signs): Change From Baseline to End of Study
Description: Orthostatic blood pressure was measured after the participant had been supine (lying down with their face up) for at least 5 minutes and then, after the participant had been standing for 2 minutes. When vital sign measurements were scheduled at the same time as a blood collection, vital sign measurements were obtained prior to blood collection.
Time Frame: Baseline, Weeks 1, 6, 26, and 52 (orthostatic and standing); Baseline, Weeks 2, 4, 13, and 39 (supine)
Population: Safety Analysis Set: all participants who received any ABBV-951 infusion with available data
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | ABBV-951 Low Dose Subgroup | ABBV-951 High Dose Subgroup | ABBV-951 All Participants
Number analyzed (Participants) | 128 | 112 | 240
mmHg
  Week 1- orthostatic: number analyzed (Participants) | 119 | 106 | 225
  Week 1- orthostatic | -1.5 (12.00) | 3.5 (16.01) | 0.9 (14.22)
  Week 6- orthostatic: number analyzed (Participants) | 97 | 89 | 186
  Week 6- orthostatic | -1.5 (11.85) | 2.6 (17.33) | 0.5 (14.83)
  Week 26- orthostatic: number analyzed (Participants) | 69 | 61 | 130
  Week 26- orthostatic | -2.4 (16.25) | -0.3 (14.38) | -1.4 (15.38)
  Week 52- orthostatic: number analyzed (Participants) | 70 | 58 | 128
  Week 52- orthostatic | -1.3 (14.59) | 0.7 (13.75) | -0.4 (14.19)
  Week 1- standing: number analyzed (Participants) | 122 | 106 | 228
  Week 1- standing | -2.3 (17.05) | -1.3 (25.50) | -1.9 (21.35)
  Week 6- standing: number analyzed (Participants) | 99 | 90 | 189
  Week 6- standing | -2.9 (18.32) | -3.1 (25.89) | -3.0 (22.19)
  Week 26- standing: number analyzed (Participants) | 71 | 61 | 132
  Week 26- standing | -4.7 (19.23) | -4.0 (21.01) | -4.4 (20.00)
  Week 52- standing: number analyzed (Participants) | 72 | 58 | 130
  Week 52- standing | -3.9 (19.81) | -1.5 (20.91) | -2.8 (20.26)
  Week 2- supine: number analyzed (Participants) | 121 | 109 | 230
  Week 2- supine | -1.0 (16.75) | -4.5 (21.94) | -2.7 (19.42)
  Week 4- supine: number analyzed (Participants) | 99 | 89 | 188
  Week 4- supine | -1.2 (16.67) | -6.7 (22.99) | -3.8 (20.05)
  Week 13- supine: number analyzed (Participants) | 29 | 17 | 46
  Week 13- supine | -4.0 (18.34) | -1.8 (24.89) | -3.2 (20.75)
  Week 39- supine: number analyzed (Participants) | 77 | 66 | 143
  Week 39- supine | -1.7 (19.12) | -1.8 (22.08) | -1.7 (20.47)

42. Primary Outcome: Orthostatic Diastolic Blood Pressure (Vital Signs): Change From Baseline to End of Study
Description: as for outcome 41
Time Frame: Baseline, Weeks 1, 6, 26, and 52 (orthostatic and standing); Baseline, Weeks 2, 4, 13, and 39 (supine)
Population: Safety Analysis Set: all participants who received any ABBV-951 infusion with available data
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | ABBV-951 Low Dose Subgroup | ABBV-951 High Dose Subgroup | ABBV-951 All Participants
Number analyzed (Participants) | 128 | 112 | 240
mmHg
  Week 1- orthostatic: number analyzed (Participants) | 119 | 106 | 225
  Week 1- orthostatic | -1.9 (10.61) | -0.7 (13.27) | -1.3 (11.92)
  Week 6- orthostatic: number analyzed (Participants) | 97 | 89 | 186
  Week 6- orthostatic | 0.0 (10.91) | -0.6 (10.00) | -0.3 (10.46)
  Week 26- orthostatic: number analyzed (Participants) | 69 | 61 | 130
  Week 26- orthostatic | -1.7 (12.99) | 0.3 (10.16) | -0.7 (11.75)
  Week 52- orthostatic: number analyzed (Participants) | 70 | 58 | 128
  Week 52- orthostatic | -1.5 (10.44) | 0.8 (11.42) | -0.4 (10.91)
  Week 1- standing: number analyzed (Participants) | 122 | 106 | 228
  Week 1- standing | -2.6 (12.00) | -2.1 (13.87) | -2.4 (12.88)
  Week 6- standing: number analyzed (Participants) | 99 | 90 | 189
  Week 6- standing | -0.8 (12.27) | -2.2 (14.76) | -1.5 (13.50)
  Week 26- standing: number analyzed (Participants) | 71 | 61 | 132
  Week 26- standing | -4.0 (12.20) | -1.2 (14.67) | -2.7 (13.42)
  Week 52- standing: number analyzed (Participants) | 72 | 58 | 130
  Week 52- standing | -1.7 (12.55) | 1.1 (12.01) | -0.4 (12.34)
  Week 2- supine: number analyzed (Participants) | 121 | 109 | 230
  Week 2- supine | -1.1 (12.46) | -1.3 (13.46) | -1.2 (12.91)
  Week 4- supine: number analyzed (Participants) | 99 | 89 | 188
  Week 4- supine | -1.4 (12.06) | -2.1 (12.80) | -1.7 (12.38)
  Week 13- supine: number analyzed (Participants) | 29 | 17 | 46
  Week 13- supine | -2.6 (12.52) | -0.5 (9.59) | -1.8 (11.46)
  Week 39- supine: number analyzed (Participants) | 77 | 66 | 143
  Week 39- supine | 0.2 (12.16) | 0.2 (12.77) | 0.2 (12.40)

43. Primary Outcome: Orthostatic Pulse Rate (Vital Signs): Change From Baseline to End of Study
Description: Orthostatic pulse rate was measured after the participant had been supine (lying down with their face up) for at least 5 minutes and then, after the participant had been standing for 2 minutes. When vital sign measurements were scheduled at the same time as a blood collection, vital sign measurements were obtained prior to blood collection.
Time Frame: Baseline, Weeks 1, 6, 26, and 52 (orthostatic and standing); Baseline, Weeks 2, 4, 13, and 39 (supine)
Population: Safety Analysis Set: all participants who received any ABBV-951 infusion with available data
Measure: Mean (Standard Deviation); unit: beats/minute
Arm/Group | ABBV-951 Low Dose Subgroup | ABBV-951 High Dose Subgroup | ABBV-951 All Participants
Number analyzed (Participants) | 128 | 112 | 240
beats/minute
  Week 1- orthostatic: number analyzed (Participants) | 119 | 106 | 225
  Week 1- orthostatic | -1.5 (8.49) | -1.8 (10.49) | -1.6 (9.46)
  Week 6- orthostatic: number analyzed (Participants) | 97 | 89 | 186
  Week 6- orthostatic | -0.5 (10.86) | 0.2 (10.16) | -0.1 (10.51)
  Week 26- orthostatic: number analyzed (Participants) | 69 | 61 | 130
  Week 26- orthostatic | -0.9 (8.90) | 0.3 (9.32) | -0.4 (9.08)
  Week 52- orthostatic: number analyzed (Participants) | 70 | 58 | 128
  Week 52- orthostatic | 0.5 (9.72) | -0.5 (8.55) | 0.0 (9.19)
  Week 1- standing: number analyzed (Participants) | 122 | 106 | 228
  Week 1- standing | -5.1 (11.43) | -2.6 (12.50) | -3.9 (11.98)
  Week 6- standing: number analyzed (Participants) | 99 | 90 | 189
  Week 6- standing | -3.1 (12.45) | -3.0 (12.23) | -3.1 (12.31)
  Week 26- standing: number analyzed (Participants) | 71 | 61 | 132
  Week 26- standing | -2.9 (12.29) | -2.4 (12.43) | -2.7 (12.31)
  Week 52- standing: number analyzed (Participants) | 72 | 58 | 130
  Week 52- standing | -3.8 (12.88) | -4.3 (11.56) | -4.0 (12.27)
  Week 2- supine: number analyzed (Participants) | 121 | 109 | 230
  Week 2- supine | -3.3 (10.05) | -0.6 (11.10) | -2.0 (10.62)
  Week 4- supine: number analyzed (Participants) | 99 | 89 | 188
  Week 4- supine | -2.6 (10.06) | -3.3 (12.60) | -3.0 (11.31)
  Week 13- supine: number analyzed (Participants) | 29 | 17 | 46
  Week 13- supine | 1.1 (11.72) | -4.8 (7.60) | -1.1 (10.68)
  Week 39- supine: number analyzed (Participants) | 77 | 66 | 143
  Week 39- supine | -3.7 (11.76) | -3.2 (11.16) | -3.4 (11.45)

44. Primary Outcome: Electrocardiogram (ECG) Mean Heart Rate: Change From Baseline to End of Study
Description: 12-lead electrocardiograms (ECGs) were recorded at study visits after the participant had been supine for at least 5 minutes. Participants were instructed to remain stationary (no talking, laughing, deep breathing, sleeping, or swallowing) for approximately 10 seconds during the ECG recording. When an ECG was recorded at a time near that of a blood collection, the ECG was obtained prior to the blood collection. ECGs on Day 1 were recorded after initiation of the continuous subcutaneous infusion (CSCI) of ABBV-951 prior to the end of the study visit.
Time Frame: Baseline, Day 1 (postdose), Weeks 6 and 52
Population: Safety Analysis Set: all participants who received any ABBV-951 infusion with available data
Measure: Mean (Standard Deviation); unit: beats/minute
Arm/Group | ABBV-951 Low Dose Subgroup | ABBV-951 High Dose Subgroup | ABBV-951 All Participants
Number analyzed (Participants) | 131 | 113 | 244
beats/minute
  Day 1 (postdose): number analyzed (Participants) | 126 | 111 | 237
  Day 1 (postdose) | 2.1 (9.51) | 2.2 (9.76) | 2.1 (9.61)
  Week 6: number analyzed (Participants) | 100 | 88 | 188
  Week 6 | -2.3 (8.60) | -2.2 (10.28) | -2.2 (9.40)
  Week 52: number analyzed (Participants) | 73 | 58 | 131
  Week 52 | -3.7 (9.51) | -0.7 (11.36) | -2.3 (10.44)

45. Primary Outcome: Electrocardiogram (ECG) Aggregate PR Interval: Change From Baseline to End of Study
Description: as for outcome 44
Time Frame: Baseline, Day 1 (postdose), Weeks 6 and 52
Population: Safety Analysis Set: all participants who received any ABBV-951 infusion with available data
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | ABBV-951 Low Dose Subgroup | ABBV-951 High Dose Subgroup | ABBV-951 All Participants
Number analyzed (Participants) | 130 | 107 | 237
milliseconds
  Day 1 (postdose): number analyzed (Participants) | 125 | 105 | 230
  Day 1 (postdose) | 0.4 (14.08) | -0.1 (13.76) | 0.2 (13.91)
  Week 6: number analyzed (Participants) | 99 | 84 | 183
  Week 6 | 0.5 (13.97) | 1.1 (16.84) | 0.8 (15.31)
  Week 52: number analyzed (Participants) | 72 | 54 | 126
  Week 52 | 1.5 (12.48) | -5.8 (20.54) | -1.6 (16.75)

46. Primary Outcome: Electrocardiogram (ECG) Aggregate QRS Duration: Change From Baseline to End of Study
Description: as for outcome 44
Time Frame: Baseline, Day 1 (postdose), Weeks 6 and 52
Population: Safety Analysis Set: all participants who received any ABBV-951 infusion with available data
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | ABBV-951 Low Dose Subgroup | ABBV-951 High Dose Subgroup | ABBV-951 All Participants
Number analyzed (Participants) | 131 | 113 | 244
milliseconds
  Day 1 (postdose): number analyzed (Participants) | 126 | 111 | 237
  Day 1 (postdose) | -2.3 (7.32) | -0.8 (8.41) | -1.6 (7.87)
  Week 6: number analyzed (Participants) | 100 | 88 | 188
  Week 6 | -0.5 (8.32) | 1.6 (8.96) | 0.5 (8.67)
  Week 52: number analyzed (Participants) | 72 | 58 | 130
  Week 52 | -0.2 (6.85) | 0.9 (7.29) | 0.3 (7.04)

47. Primary Outcome: Electrocardiogram (ECG) Aggregate QT Interval: Change From Baseline to End of Study
Description: as for outcome 44
Time Frame: Baseline, Day 1 (postdose), Weeks 6 and 52
Population: Safety Analysis Set: all participants who received any ABBV-951 infusion with available data
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | ABBV-951 Low Dose Subgroup | ABBV-951 High Dose Subgroup | ABBV-951 All Participants
Number analyzed (Participants) | 131 | 113 | 244
milliseconds
  Day 1 (postdose): number analyzed (Participants) | 126 | 111 | 237
  Day 1 (postdose) | -5.3 (20.72) | -4.2 (23.99) | -4.8 (22.27)
  Week 6: number analyzed (Participants) | 99 | 88 | 187
  Week 6 | 6.4 (20.96) | 6.4 (24.61) | 6.4 (22.69)
  Week 52: number analyzed (Participants) | 72 | 58 | 130
  Week 52 | 9.8 (24.66) | 4.3 (26.24) | 7.3 (25.42)

48. Primary Outcome: Electrocardiogram (ECG) Aggregate QTcB Interval: Change From Baseline to End of Study
Description: as for outcome 44
Time Frame: Baseline, Day 1 (postdose), Weeks 6 and 52
Population: Safety Analysis Set: all participants who received any ABBV-951 infusion with available data
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | ABBV-951 Low Dose Subgroup | ABBV-951 High Dose Subgroup | ABBV-951 All Participants
Number analyzed (Participants) | 131 | 113 | 244
milliseconds
  Day 1 (postdose): number analyzed (Participants) | 126 | 111 | 237
  Day 1 (postdose) | 1.2 (17.96) | 2.0 (17.21) | 1.6 (17.58)
  Week 6: number analyzed (Participants) | 99 | 88 | 187
  Week 6 | 1.0 (19.91) | 0.6 (18.34) | 0.8 (19.14)
  Week 52: number analyzed (Participants) | 72 | 58 | 130
  Week 52 | -0.1 (20.84) | 2.1 (18.33) | 0.9 (19.72)

49. Primary Outcome: Electrocardiogram (ECG) Aggregate QTcF Interval: Change From Baseline to End of Study
Description: as for outcome 44
Time Frame: Baseline, Day 1 (postdose), Weeks 6 and 52
Population: Safety Analysis Set: all participants who received any ABBV-951 infusion with available data
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | ABBV-951 Low Dose Subgroup | ABBV-951 High Dose Subgroup | ABBV-951 All Participants
Number analyzed (Participants) | 131 | 113 | 244
milliseconds
  Day 1 (postdose): number analyzed (Participants) | 126 | 111 | 237
  Day 1 (postdose) | -1.0 (14.03) | -0.2 (15.75) | -0.6 (14.84)
  Week 6: number analyzed (Participants) | 99 | 88 | 187
  Week 6 | 3.1 (16.49) | 2.6 (15.63) | 2.9 (16.05)
  Week 52: number analyzed (Participants) | 72 | 58 | 130
  Week 52 | 3.4 (18.05) | 2.9 (15.40) | 3.2 (16.86)

50. Primary Outcome: Electrocardiogram (ECG) Aggregate RR Interval: Change From Baseline to End of Study
Description: as for outcome 44
Time Frame: Baseline, Day 1 (postdose), Weeks 6 and 52
Population: Safety Analysis Set: all participants who received any ABBV-951 infusion with available data
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | ABBV-951 Low Dose Subgroup | ABBV-951 High Dose Subgroup | ABBV-951 All Participants
Number analyzed (Participants) | 131 | 113 | 244
milliseconds
  Day 1 (postdose): number analyzed (Participants) | 126 | 111 | 237
  Day 1 (postdose) | -30.7 (122.48) | -28.3 (113.02) | -29.6 (117.90)
  Week 6: number analyzed (Participants) | 100 | 88 | 188
  Week 6 | 22.6 (112.51) | 26.1 (129.35) | 24.2 (120.37)
  Week 52: number analyzed (Participants) | 73 | 58 | 131
  Week 52 | 41.8 (122.96) | 9.4 (141.91) | 27.5 (132.15)

51. Secondary Outcome: Average Daily Normalized "Off" Time: Change From Baseline to End of Study
Description: Upon awakening and every 30 minutes during their normal waking time, participants recorded their state in the Parkinson's Disease Diary (PD Diary) for 2 consecutive days prior to study visits.
  "Off" time is defined as periods of poor mobility, tremor, slowness, and stiffness. The daily "On" and "Off" times were normalized to a typical waking day (16 hours) to account for different sleep patterns across participants. When "Off" was the first morning symptom upon awakening, this was considered morning akinesia in this study.
  Baseline value is defined as the average of normalized "Off" time collected over the 2 PD Diary days before the Enrollment visit. Negative changes from Baseline indicate improvement.
Time Frame: Baseline, Weeks 1, 6, 13, 26, 39, and 52
Population: Full Analysis Set: all participants who received any ABBV-951 infusion and had a Baseline and treatment observation for at least 1 efficacy outcome measure
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | ABBV-951 Low Dose Subgroup | ABBV-951 High Dose Subgroup | ABBV-951 All Participants
Number analyzed (Participants) | 126 | 110 | 236
hours
  Week 1: number analyzed (Participants) | 120 | 105 | 225
  Week 1 | -2.04 (3.51) | -1.84 (3.88) | -1.95 (3.68)
  Week 6: number analyzed (Participants) | 110 | 95 | 205
  Week 6 | -2.43 (3.66) | -2.36 (3.56) | -2.40 (3.61)
  Week 13: number analyzed (Participants) | 63 | 51 | 114
  Week 13 | -2.50 (3.83) | -2.34 (3.57) | -2.43 (3.70)
  Week 26: number analyzed (Participants) | 69 | 62 | 131
  Week 26 | -3.31 (3.36) | -3.38 (3.15) | -3.35 (3.25)
  Week 39: number analyzed (Participants) | 68 | 54 | 122
  Week 39 | -3.25 (3.43) | -3.52 (2.92) | -3.37 (3.21)
  Week 52: number analyzed (Participants) | 62 | 54 | 116
  Week 52 | -3.43 (3.16) | -3.59 (3.11) | -3.51 (3.12)
Statistical Analysis 1: Comparison: ABBV-951 Low Dose Subgroup; Week 1 vs Baseline; Test type: Superiority — A paired-sample t-test was performed to test the change from Baseline; p < 0.001, paired-sample t-test
Statistical Analysis 2: Comparison: ABBV-951 High Dose Subgroup; Week 1 vs Baseline; Test type: Superiority — A paired-sample t-test was performed to test the change from Baseline; p < 0.001, paired-sample t-test
Statistical Analysis 3: Comparison: ABBV-951 All Participants; Week 1 vs Baseline; Test type: Superiority — A paired-sample t-test was performed to test the change from Baseline; p < 0.001, paired-sample t-test
Statistical Analysis 4: Comparison: ABBV-951 Low Dose Subgroup; Week 6 vs Baseline; Test type: Superiority — A paired-sample t-test was performed to test the change from Baseline; p < 0.001, paired-sample t-test
Statistical Analysis 5: Comparison: ABBV-951 High Dose Subgroup; Week 6 vs Baseline; Test type: Superiority — A paired-sample t-test was performed to test the change from Baseline; p < 0.001, paired-sample t-test
Statistical Analysis 6: Comparison: ABBV-951 All Participants; Week 6 vs Baseline; Test type: Superiority — A paired-sample t-test was performed to test the change from Baseline; p < 0.001, paired-sample t-test
Statistical Analysis 7: Comparison: ABBV-951 Low Dose Subgroup; Week 13 vs Baseline; Test type: Superiority — A paired-sample t-test was performed to test the change from Baseline; p < 0.001, paired-sample t-test
Statistical Analysis 8: Comparison: ABBV-951 High Dose Subgroup; Week 13 vs Baseline; Test type: Superiority — A paired-sample t-test was performed to test the change from Baseline; p < 0.001, paired-sample t-test
Statistical Analysis 9: Comparison: ABBV-951 All Participants; Week 13 vs Baseline; Test type: Superiority — A paired-sample t-test was performed to test the change from Baseline; p < 0.001, paired-sample t-test
Statistical Analysis 10: Comparison: ABBV-951 Low Dose Subgroup; Week 26 vs Baseline; Test type: Superiority — A paired-sample t-test was performed to test the change from Baseline; p < 0.001, paired-sample t-test
Statistical Analysis 11: Comparison: ABBV-951 High Dose Subgroup; Week 26 vs Baseline; Test type: Superiority — A paired-sample t-test was performed to test the change from Baseline; p < 0.001, paired-sample t-test
Statistical Analysis 12: Comparison: ABBV-951 All Participants; Week 26 vs Baseline; Test type: Superiority — Week 26 vs Baseline; p < 0.001, paired-sample t-test
Statistical Analysis 13: Comparison: ABBV-951 Low Dose Subgroup; Week 39 vs Baseline; Test type: Superiority — A paired-sample t-test was performed to test the change from Baseline; p < 0.001, paired-sample t-test
Statistical Analysis 14: Comparison: ABBV-951 High Dose Subgroup; Week 39 vs Baseline; Test type: Superiority — A paired-sample t-test was performed to test the change from Baseline; p < 0.001, paired-sample t-test
Statistical Analysis 15: Comparison: ABBV-951 All Participants; Week 39 vs Baseline; Test type: Superiority — A paired-sample t-test was performed to test the change from Baseline; p < 0.001, paired-sample t-test
Statistical Analysis 16: Comparison: ABBV-951 Low Dose Subgroup; Week 52 vs Baseline; Test type: Superiority — A paired-sample t-test was performed to test the change from Baseline; p < 0.001, paired-sample t-test
Statistical Analysis 17: Comparison: ABBV-951 High Dose Subgroup; Week 52 vs Baseline; Test type: Superiority — A paired-sample t-test was performed to test the change from Baseline; p < 0.001, paired-sample t-test
Statistical Analysis 18: Comparison: ABBV-951 All Participants; Week 52 vs Baseline; Test type: Superiority — A paired-sample t-test was performed to test the change from Baseline; p < 0.001, paired-sample t-test

52. Secondary Outcome: Average Daily Normalized "On" Time With Troublesome Dyskinesia: Change From Baseline to End of Study
Description: Upon awakening and every 30 minutes during their normal waking time, participants recorded their state in the Parkinson's Disease Diary (PD Diary) for 2 consecutive days prior to study visits.
  "On" time is defined as periods of good motor symptom control. The daily "On" and "Off" times were normalized to a typical waking day (16 hours) to account for different sleep patterns across participants.
  Baseline value is defined as the average of normalized "On" time with troublesome dyskinesia collected over the 2 PD Diary days before the Enrollment visit. Negative changes from Baseline indicate improvement.
Time Frame: Baseline, Weeks 1, 6, 13, 26, 39, and 52
Population: as for outcome 51
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | ABBV-951 Low Dose Subgroup | ABBV-951 High Dose Subgroup | ABBV-951 All Participants
Number analyzed (Participants) | 126 | 110 | 236
hours
  Week 1: number analyzed (Participants) | 120 | 105 | 225
  Week 1 | -0.00 (2.10) | 0.11 (1.64) | 0.05 (1.89)
  Week 6: number analyzed (Participants) | 110 | 95 | 205
  Week 6 | -0.56 (1.95) | -0.23 (1.05) | -0.41 (1.60)
  Week 13: number analyzed (Participants) | 63 | 51 | 114
  Week 13 | -0.60 (1.72) | -0.38 (1.04) | -0.50 (1.45)
  Week 26: number analyzed (Participants) | 69 | 62 | 131
  Week 26 | -0.61 (1.95) | -0.27 (1.73) | -0.45 (1.85)
  Week 39: number analyzed (Participants) | 68 | 54 | 122
  Week 39 | -0.49 (1.07) | -0.17 (1.59) | -0.35 (1.33)
  Week 52: number analyzed (Participants) | 62 | 54 | 116
  Week 52 | -0.64 (1.73) | 0.17 (2.53) | -0.27 (2.16)
Statistical Analysis 1: Comparison: ABBV-951 Low Dose Subgroup; Week 1 vs Baseline; Test type: Superiority — A paired-sample t-test was performed to test the change from Baseline; p > 0.999, paired-sample t-test
Statistical Analysis 2: Comparison: ABBV-951 High Dose Subgroup; Week 1 vs Baseline; Test type: Superiority — A paired-sample t-test was performed to test the change from Baseline; p = 0.5095, paired-sample t-test
Statistical Analysis 3: Comparison: ABBV-951 All Participants; Week 1 vs Baseline; Test type: Superiority — A paired-sample t-test was performed to test the change from Baseline; p = 0.6962, paired-sample t-test
Statistical Analysis 4: Comparison: ABBV-951 Low Dose Subgroup; Week 6 vs Baseline; Test type: Superiority — A paired-sample t-test was performed to test the change from Baseline; p = 0.0035, paired-sample t-test
Statistical Analysis 5: Comparison: ABBV-951 High Dose Subgroup; Week 6 vs Baseline; Test type: Superiority — A paired-sample t-test was performed to test the change from Baseline; p = 0.0324, paired-sample t-test
Statistical Analysis 6: Comparison: ABBV-951 All Participants; Week 6 vs Baseline; Test type: Superiority — A paired-sample t-test was performed to test the change from Baseline; p < 0.001, paired-sample t-test
Statistical Analysis 7: Comparison: ABBV-951 Low Dose Subgroup; Week 13 vs Baseline; Test type: Superiority — A paired-sample t-test was performed to test the change from Baseline; p = 0.0072, paired-sample t-test
Statistical Analysis 8: Comparison: ABBV-951 High Dose Subgroup; Week 13 vs Baseline; Test type: Superiority — A paired-sample t-test was performed to test the change from Baseline; p = 0.0129, paired-sample t-test
Statistical Analysis 9: Comparison: ABBV-951 All Participants; Week 13 vs Baseline; Test type: Superiority — A paired-sample t-test was performed to test the change from Baseline; p < 0.001, paired-sample t-test
Statistical Analysis 10: Comparison: ABBV-951 Low Dose Subgroup; Week 26 vs Baseline; Test type: Superiority — A paired-sample t-test was performed to test the change from Baseline; p = 0.0119, paired-sample t-test
Statistical Analysis 11: Comparison: ABBV-951 High Dose Subgroup; Week 26 vs Baseline; Test type: Superiority; p = 0.2200, paired-sample t-test — A paired-sample t-test was performed to test the change from Baseline
Statistical Analysis 12: Comparison: ABBV-951 All Participants; Week 26 vs Baseline; Test type: Superiority — A paired-sample t-test was performed to test the change from Baseline; p = 0.0063, paired-sample t-test
Statistical Analysis 13: Comparison: ABBV-951 Low Dose Subgroup; Week 39 vs Baseline; Test type: Superiority — A paired-sample t-test was performed to test the change from Baseline; p < 0.001, paired-sample t-test
Statistical Analysis 14: Comparison: ABBV-951 High Dose Subgroup; Week 39 vs Baseline; Test type: Superiority — A paired-sample t-test was performed to test the change from Baseline; p = 0.4331, paired-sample t-test
Statistical Analysis 15: Comparison: ABBV-951 All Participants; Week 39 vs Baseline; Test type: Superiority — A paired-sample t-test was performed to test the change from Baseline; p = 0.0045, paired-sample t-test
Statistical Analysis 16: Comparison: ABBV-951 Low Dose Subgroup; Week 52 vs Baseline; Test type: Superiority — A paired-sample t-test was performed to test the change from Baseline; p = 0.0049, Wilcoxon (Mann-Whitney)
Statistical Analysis 17: Comparison: ABBV-951 High Dose Subgroup; Week 52 vs Baseline; Test type: Superiority — A paired-sample t-test was performed to test the change from Baseline; p = 0.6312, paired-sample t-test
Statistical Analysis 18: Comparison: ABBV-951 All Participants; Week 52 vs Baseline; Test type: Superiority — A paired-sample t-test was performed to test the change from Baseline; p = 0.1892, paired-sample t-test

53. Secondary Outcome: Average Daily Normalized "On" Time Without Troublesome Dyskinesia: Change From Baseline to End of Study
Description: Upon awakening and every 30 minutes during their normal waking time, participants recorded their state in the Parkinson's Disease Diary (PD Diary) for 2 consecutive days prior to study visits.
  "On" time is defined as periods of good motor symptom control. The daily "On" and "Off" times were normalized to a typical waking day (16 hours) to account for different sleep patterns across participants.
  Baseline value is defined as the average of normalized "On" time without troublesome dyskinesia collected over the 2 PD Diary days before the Enrollment visit. Positive changes from Baseline indicate improvement.
Time Frame: Baseline, Weeks 1, 6, 13, 26, 39, and 52
Population: as for outcome 51
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | ABBV-951 Low Dose Subgroup | ABBV-951 High Dose Subgroup | ABBV-951 All Participants
Number analyzed (Participants) | 126 | 110 | 236
hours
  Week 1: number analyzed (Participants) | 120 | 105 | 225
  Week 1 | 2.04 (3.55) | 1.74 (4.04) | 1.90 (3.78)
  Week 6: number analyzed (Participants) | 110 | 95 | 205
  Week 6 | 2.99 (3.60) | 2.60 (3.58) | 2.81 (3.59)
  Week 13: number analyzed (Participants) | 63 | 51 | 114
  Week 13 | 3.10 (3.32) | 2.72 (3.68) | 2.93 (3.48)
  Week 26: number analyzed (Participants) | 69 | 62 | 131
  Week 26 | 3.92 (3.76) | 3.65 (3.31) | 3.79 (3.55)
  Week 39: number analyzed (Participants) | 68 | 54 | 122
  Week 39 | 3.74 (3.40) | 3.69 (3.32) | 3.71 (3.35)
  Week 52: number analyzed (Participants) | 62 | 54 | 116
  Week 52 | 4.08 (3.28) | 3.43 (3.28) | 3.77 (3.28)
Statistical Analysis 1: Comparison: ABBV-951 Low Dose Subgroup; Week 1 vs Baseline; Test type: Superiority — A paired-sample t-test was performed to test the change from Baseline; p < 0.001, paired-sample t-test
Statistical Analysis 2: Comparison: ABBV-951 High Dose Subgroup; Week 1 vs Baseline; Test type: Superiority — A paired-sample t-test was performed to test the change from Baseline; p < 0.001, paired-sample t-test
Statistical Analysis 3: Comparison: ABBV-951 All Participants; Week 1 vs Baseline; Test type: Superiority — A paired-sample t-test was performed to test the change from Baseline; p < 0.001, paired-sample t-test
Statistical Analysis 4: Comparison: ABBV-951 Low Dose Subgroup; Week 6 vs Baseline; Test type: Superiority — A paired-sample t-test was performed to test the change from Baseline; p < 0.001, paired-sample t-test
Statistical Analysis 5: Comparison: ABBV-951 High Dose Subgroup; Week 6 vs Baseline; Test type: Superiority — A paired-sample t-test was performed to test the change from Baseline; p < 0.001, paired-sample t-test
Statistical Analysis 6: Comparison: ABBV-951 All Participants; Week 6 vs Baseline; Test type: Superiority — A paired-sample t-test was performed to test the change from Baseline; p < 0.001, paired-sample t-test
Statistical Analysis 7: Comparison: ABBV-951 Low Dose Subgroup; Week 13 vs Baseline; Test type: Superiority — A paired-sample t-test was performed to test the change from Baseline; p < 0.001, paired-sample t-test
Statistical Analysis 8: Comparison: ABBV-951 High Dose Subgroup; Week 13 vs Baseline; Test type: Superiority — A paired-sample t-test was performed to test the change from Baseline; p < 0.001, paired-sample t-test
Statistical Analysis 9: Comparison: ABBV-951 All Participants; Week 13 vs Baseline; Test type: Superiority — A paired-sample t-test was performed to test the change from Baseline; p < 0.001, paired-sample t-test
Statistical Analysis 10: Comparison: ABBV-951 Low Dose Subgroup; Week 26 vs Baseline; Test type: Superiority — A paired-sample t-test was performed to test the change from Baseline; p < 0.001, paired-sample t-test
Statistical Analysis 11: Comparison: ABBV-951 High Dose Subgroup; Week 26 vs Baseline; Test type: Superiority — A paired-sample t-test was performed to test the change from Baseline; p < 0.001, paired-sample t-test
Statistical Analysis 12: Comparison: ABBV-951 All Participants; Week 26 vs Baseline; Test type: Superiority — A paired-sample t-test was performed to test the change from Baseline; p < 0.001, paired-sample t-test
Statistical Analysis 13: Comparison: ABBV-951 Low Dose Subgroup; Week 39 vs Baseline; Test type: Superiority — A paired-sample t-test was performed to test the change from Baseline; p < 0.001, paired-sample t-test
Statistical Analysis 14: Comparison: ABBV-951 High Dose Subgroup; Week 39 vs Baseline; Test type: Superiority — A paired-sample t-test was performed to test the change from Baseline; p < 0.001, paired-sample t-test
Statistical Analysis 15: Comparison: ABBV-951 All Participants; Week 39 vs Baseline; Test type: Superiority — A paired-sample t-test was performed to test the change from Baseline; p < 0.001, paired-sample t-test
Statistical Analysis 16: Comparison: ABBV-951 Low Dose Subgroup; Week 52 vs Baseline; Test type: Superiority — A paired-sample t-test was performed to test the change from Baseline; p < 0.001, paired-sample t-test
Statistical Analysis 17: Comparison: ABBV-951 High Dose Subgroup; Week 52 vs Baseline; Test type: Superiority — A paired-sample t-test was performed to test the change from Baseline; p < 0.001, paired-sample t-test
Statistical Analysis 18: Comparison: ABBV-951 All Participants; Week 52 vs Baseline; Test type: Superiority — A paired-sample t-test was performed to test the change from Baseline; p < 0.001, paired-sample t-test

54. Secondary Outcome: Movement Disorder Society-Unified Parkinson's Disease Rating Scale (MDS-UPDRS) Part I Score: Change From Baseline to End of Study
Description: The Movement Disorder Society-Unified Parkinson's Disease Rating Scale (MDS-UPDRS) is an investigator-used rating tool to follow the longitudinal course of Parkinson's Disease (PD). Part I assesses the participant's non-motor aspects of experiences of daily living (nM-EDL) with 13 questions. (The numeric score for each question is between 0-4; 0=Normal,1=Slight,2=Mild,3=Moderate,4=Severe). Part I scores range from 0 to 52, with higher scores indicating more severe symptoms of PD. Negative changes from Baseline indicate improvement.
Time Frame: Baseline, Day 2, Weeks 1, 2, 3, 4, 6, 13, 26, 39, and 52
Population: as for outcome 51
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ABBV-951 Low Dose Subgroup | ABBV-951 High Dose Subgroup | ABBV-951 All Participants
Number analyzed (Participants) | 131 | 113 | 244
units on a scale
  Day 2: number analyzed (Participants) | 120 | 102 | 222
  Day 2 | -2.6 (4.28) | -1.8 (3.61) | -2.3 (4.00)
  Week 1: number analyzed (Participants) | 120 | 106 | 226
  Week 1 | -2.6 (5.84) | -3.3 (5.50) | -2.9 (5.68)
  Week 2: number analyzed (Participants) | 117 | 95 | 212
  Week 2 | -2.5 (5.29) | -2.1 (5.10) | -2.3 (5.20)
  Week 3: number analyzed (Participants) | 107 | 96 | 203
  Week 3 | -2.3 (5.65) | -2.9 (5.91) | -2.6 (5.77)
  Week 4: number analyzed (Participants) | 109 | 94 | 203
  Week 4 | -1.7 (6.22) | -3.0 (5.42) | -2.3 (5.88)
  Week 6: number analyzed (Participants) | 104 | 89 | 193
  Week 6 | -1.1 (7.00) | -1.7 (5.15) | -1.4 (6.21)
  Week 13: number analyzed (Participants) | 93 | 77 | 170
  Week 13 | -1.8 (5.80) | -1.7 (5.59) | -1.7 (5.69)
  Week 26: number analyzed (Participants) | 79 | 69 | 148
  Week 26 | -1.1 (5.01) | -0.7 (5.88) | -0.9 (5.42)
  Week 39: number analyzed (Participants) | 75 | 60 | 135
  Week 39 | -0.7 (5.64) | 0.1 (6.00) | -0.4 (5.80)
  Week 52: number analyzed (Participants) | 75 | 58 | 133
  Week 52 | -0.5 (5.30) | -1.3 (6.22) | -0.9 (5.71)
Statistical Analysis 1: Comparison: ABBV-951 Low Dose Subgroup; Day 2 vs Baseline; Test type: Superiority — A paired-sample t-test was performed to test the change from Baseline; p < 0.001, paired-sample t-test
Statistical Analysis 2: Comparison: ABBV-951 High Dose Subgroup; Day 2 vs Baseline; Test type: Superiority — A paired-sample t-test was performed to test the change from Baseline; p < 0.001, paired-sample t-test
Statistical Analysis 3: Comparison: ABBV-951 All Participants; Day 2 vs Baseline; Test type: Superiority — A paired-sample t-test was performed to test the change from Baseline; p < 0.001, paired-sample t-test
Statistical Analysis 4: Comparison: ABBV-951 Low Dose Subgroup; Week 1 vs Baseline; Test type: Superiority — A paired-sample t-test was performed to test the change from Baseline; p < 0.001, paired-sample t-test
Statistical Analysis 5: Comparison: ABBV-951 High Dose Subgroup; Week 1 vs Baseline; Test type: Superiority — A paired-sample t-test was performed to test the change from Baseline; p < 0.001, paired-sample t-test
Statistical Analysis 6: Comparison: ABBV-951 All Participants; Week 1 vs Baseline; Test type: Superiority — A paired-sample t-test was performed to test the change from Baseline; p < 0.001, paired-sample t-test
Statistical Analysis 7: Comparison: ABBV-951 Low Dose Subgroup; Week 2 vs Baseline; Test type: Superiority — A paired-sample t-test was performed to test the change from Baseline; p < 0.001, paired-sample t-test
Statistical Analysis 8: Comparison: ABBV-951 High Dose Subgroup; Week 2 vs Baseline; Test type: Superiority — A paired-sample t-test was performed to test the change from Baseline; p < 0.001, paired-sample t-test
Statistical Analysis 9: Comparison: ABBV-951 All Participants; Week 2 vs Baseline; Test type: Superiority — A paired-sample t-test was performed to test the change from Baseline; p < 0.001, paired-sample t-test
Statistical Analysis 10: Comparison: ABBV-951 Low Dose Subgroup; Week 3 vs Baseline; Test type: Superiority — A paired-sample t-test was performed to test the change from Baseline; p < 0.001, paired-sample t-test
Statistical Analysis 11: Comparison: ABBV-951 High Dose Subgroup; Week 3 vs Baseline; Test type: Superiority — A paired-sample t-test was performed to test the change from Baseline; p < 0.001, paired-sample t-test
Statistical Analysis 12: Comparison: ABBV-951 All Participants; Week 3 vs Baseline; Test type: Superiority — A paired-sample t-test was performed to test the change from Baseline; p < 0.001, paired-sample t-test
Statistical Analysis 13: Comparison: ABBV-951 Low Dose Subgroup; Week 4 vs Baseline; Test type: Superiority — A paired-sample t-test was performed to test the change from Baseline; p = 0.0042, paired-sample t-test
Statistical Analysis 14: Comparison: ABBV-951 High Dose Subgroup; Week 4 vs Baseline; Test type: Superiority — A paired-sample t-test was performed to test the change from Baseline; p < 0.001, paired-sample t-test
Statistical Analysis 15: Comparison: ABBV-951 All Participants; Week 4 vs Baseline; Test type: Superiority — A paired-sample t-test was performed to test the change from Baseline; p < 0.001, paired-sample t-test
Statistical Analysis 16: Comparison: ABBV-951 Low Dose Subgroup; Week 6 vs Baseline; Test type: Superiority — A paired-sample t-test was performed to test the change from Baseline; p = 0.1135, paired-sample t-test
Statistical Analysis 17: Comparison: ABBV-951 High Dose Subgroup; Week 6 vs Baseline; Test type: Superiority — A paired-sample t-test was performed to test the change from Baseline; p = 0.0029, paired-sample t-test
Statistical Analysis 18: Comparison: ABBV-951 All Participants; Week 6 vs Baseline; Test type: Superiority — A paired-sample t-test was performed to test the change from Baseline; p = 0.0026, paired-sample t-test
Statistical Analysis 19: Comparison: ABBV-951 Low Dose Subgroup; Week 13 vs Baseline; Test type: Superiority — A paired-sample t-test was performed to test the change from Baseline; p = 0.0034, paired-sample t-test
Statistical Analysis 20: Comparison: ABBV-951 High Dose Subgroup; Week 13 vs Baseline; Test type: Superiority — A paired-sample t-test was performed to test the change from Baseline; p = 0.0103, paired-sample t-test
Statistical Analysis 21: Comparison: ABBV-951 All Participants; Week 13 vs Baseline; Test type: Superiority — A paired-sample t-test was performed to test the change from Baseline; p < 0.001, paired-sample t-test
Statistical Analysis 22: Comparison: ABBV-951 Low Dose Subgroup; Week 26 vs Baseline; Test type: Superiority — A paired-sample t-test was performed to test the change from Baseline; p = 0.0493, paired-sample t-test
Statistical Analysis 23: Comparison: ABBV-951 High Dose Subgroup; Week 26 vs Baseline; Test type: Superiority — A paired-sample t-test was performed to test the change from Baseline; p = 0.3003, paired-sample t-test
Statistical Analysis 24: Comparison: ABBV-951 All Participants; Week 26 vs Baseline; Test type: Superiority — A paired-sample t-test was performed to test the change from Baseline; p = 0.0354, paired-sample t-test
Statistical Analysis 25: Comparison: ABBV-951 Low Dose Subgroup; Week 39 vs Baseline; Test type: Superiority — A paired-sample t-test was performed to test the change from Baseline; p = 0.2553, paired-sample t-test
Statistical Analysis 26: Comparison: ABBV-951 High Dose Subgroup; Week 39 vs Baseline; Test type: Superiority — A paired-sample t-test was performed to test the change from Baseline; p = 0.8640, paired-sample t-test
Statistical Analysis 27: Comparison: ABBV-951 All Participants; Week 39 vs Baseline; Test type: Superiority — A paired-sample t-test was performed to test the change from Baseline; p = 0.4774, paired-sample t-test
Statistical Analysis 28: Comparison: ABBV-951 Low Dose Subgroup; Week 52 vs Baseline; Test type: Superiority — A paired-sample t-test was performed to test the change from Baseline; p = 0.3865, paired-sample t-test
Statistical Analysis 29: Comparison: ABBV-951 High Dose Subgroup; Week 52 vs Baseline; Test type: Superiority — A paired-sample t-test was performed to test the change from Baseline; p = 0.1186, paired-sample t-test
Statistical Analysis 30: Comparison: ABBV-951 All Participants; Week 52 vs Baseline; Test type: Superiority — A paired-sample t-test was performed to test the change from Baseline; p = 0.0830, paired-sample t-test

55. Secondary Outcome: Movement Disorder Society-Unified Parkinson's Disease Rating Scale (MDS-UPDRS) Part II Score: Change From Baseline to End of Study
Description: The Movement Disorder Society-Unified Parkinson's Disease Rating Scale (MDS-UPDRS) is an investigator-used rating tool to follow the longitudinal course of Parkinson's Disease (PD). Part II assesses the participant's motor experiences of daily living (M-EDL) with 13 questions. (The numeric score for each question is between 0-4; 0=Normal,1=Slight,2=Mild,3=Moderate,4=Severe). Part II scores range from 0 to 52, with higher scores indicating more severe symptoms of PD. Negative changes from Baseline indicate improvement.
Time Frame: Baseline, Day 2, Weeks 1, 2, 3, 4, 6, 13, 26, 39, and 52
Population: as for outcome 51
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ABBV-951 Low Dose Subgroup | ABBV-951 High Dose Subgroup | ABBV-951 All Participants
Number analyzed (Participants) | 131 | 113 | 244
units on a scale
  Day 2: number analyzed (Participants) | 120 | 102 | 222
  Day 2 | -2.8 (4.55) | -1.2 (4.25) | -2.1 (4.47)
  Week 1: number analyzed (Participants) | 120 | 106 | 226
  Week 1 | -3.6 (4.98) | -3.9 (5.85) | -3.7 (5.40)
  Week 2: number analyzed (Participants) | 117 | 95 | 212
  Week 2 | -3.3 (6.06) | -3.4 (6.53) | -3.3 (6.26)
  Week 3: number analyzed (Participants) | 107 | 96 | 203
  Week 3 | -3.5 (5.83) | -3.9 (6.63) | -3.7 (6.21)
  Week 4: number analyzed (Participants) | 109 | 84 | 203
  Week 4 | -2.6 (5.50) | -4.9 (6.32) | -3.7 (5.98)
  Week 6: number analyzed (Participants) | 104 | 89 | 193
  Week 6 | -2.5 (6.60) | -4.2 (6.09) | -3.3 (6.41)
  Week 13: number analyzed (Participants) | 93 | 77 | 170
  Week 13 | -3.2 (6.44) | -4.3 (6.57) | -3.7 (6.50)
  Week 26: number analyzed (Participants) | 79 | 69 | 148
  Week 26 | -2.6 (6.27) | -3.9 (7.05) | -3.2 (6.65)
  Week 39: number analyzed (Participants) | 75 | 60 | 135
  Week 39 | -2.6 (6.32) | -4.0 (6.93) | -3.2 (6.61)
  Week 52: number analyzed (Participants) | 75 | 58 | 133
  Week 52 | -2.1 (6.94) | -4.5 (7.07) | -3.2 (7.07)
Statistical Analysis 1: Comparison: ABBV-951 Low Dose Subgroup; Day 2 vs Baseline; Test type: Superiority — A paired-sample t-test was performed to test the change from Baseline; p < 0.001, paired-sample t-test
Statistical Analysis 2: Comparison: ABBV-951 High Dose Subgroup; Day 2 vs Baseline; Test type: Superiority — A paired-sample t-test was performed to test the change from Baseline; p = 0.0041, paired-sample t-test
Statistical Analysis 3: Comparison: ABBV-951 All Participants; Day 2 vs Baseline; Test type: Superiority — A paired-sample t-test was performed to test the change from Baseline; p < 0.001, paired-sample t-test
Statistical Analysis 4: Comparison: ABBV-951 Low Dose Subgroup; Week 1 vs Baseline; Test type: Superiority — A paired-sample t-test was performed to test the change from Baseline; p < 0.001, paired-sample t-test
Statistical Analysis 5: Comparison: ABBV-951 High Dose Subgroup; Week 1 vs Baseline; Test type: Superiority — A paired-sample t-test was performed to test the change from Baseline; p < 0.001, paired-sample t-test
Statistical Analysis 6: Comparison: ABBV-951 All Participants; Week 1 vs Baseline; Test type: Superiority — A paired-sample t-test was performed to test the change from Baseline; p < 0.001, paired-sample t-test
Statistical Analysis 7: Comparison: ABBV-951 Low Dose Subgroup; Week 2 vs Baseline; Test type: Superiority — A paired-sample t-test was performed to test the change from Baseline; p < 0.001, paired-sample t-test
Statistical Analysis 8: Comparison: ABBV-951 High Dose Subgroup; Week 2 vs Baseline; Test type: Superiority — A paired-sample t-test was performed to test the change from Baseline; p < 0.001, paired-sample t-test
Statistical Analysis 9: Comparison: ABBV-951 All Participants; Week 2 vs Baseline; Test type: Superiority — A paired-sample t-test was performed to test the change from Baseline; p < 0.001, paired-sample t-test
Statistical Analysis 10: Comparison: ABBV-951 Low Dose Subgroup; Week 3 vs Baseline; Test type: Superiority — A paired-sample t-test was performed to test the change from Baseline; p < 0.001, paired-sample t-test
Statistical Analysis 11: Comparison: ABBV-951 High Dose Subgroup; Week 3 vs Baseline; Test type: Superiority — A paired-sample t-test was performed to test the change from Baseline; p < 0.001, paired-sample t-test
Statistical Analysis 12: Comparison: ABBV-951 All Participants; Week 3 vs Baseline; Test type: Superiority — A paired-sample t-test was performed to test the change from Baseline; p < 0.001, paired-sample t-test
Statistical Analysis 13: Comparison: ABBV-951 Low Dose Subgroup; Week 4 vs Baseline; Test type: Superiority — A paired-sample t-test was performed to test the change from Baseline; p < 0.001, paired-sample t-test
Statistical Analysis 14: Comparison: ABBV-951 High Dose Subgroup; Week 4 vs Baseline; Test type: Superiority — A paired-sample t-test was performed to test the change from Baseline; p < 0.001, paired-sample t-test
Statistical Analysis 15: Comparison: ABBV-951 All Participants; Week 4 vs Baseline; Test type: Superiority — A paired-sample t-test was performed to test the change from Baseline; p < 0.001, paired-sample t-test
Statistical Analysis 16: Comparison: ABBV-951 Low Dose Subgroup; Week 6 vs Baseline; Test type: Superiority — A paired-sample t-test was performed to test the change from Baseline; p < 0.001, paired-sample t-test
Statistical Analysis 17: Comparison: ABBV-951 High Dose Subgroup; Week 6 vs Baseline; Test type: Superiority — A paired-sample t-test was performed to test the change from Baseline; p < 0.001, paired-sample t-test
Statistical Analysis 18: Comparison: ABBV-951 All Participants; Week 6 vs Baseline; Test type: Superiority — A paired-sample t-test was performed to test the change from Baseline; p < 0.001, paired-sample t-test
Statistical Analysis 19: Comparison: ABBV-951 Low Dose Subgroup; Week 13 vs Baseline; Test type: Superiority — A paired-sample t-test was performed to test the change from Baseline; p < 0.001, paired-sample t-test
Statistical Analysis 20: Comparison: ABBV-951 High Dose Subgroup; Week 13 vs Baseline; Test type: Superiority — A paired-sample t-test was performed to test the change from Baseline; p < 0.001, paired-sample t-test
Statistical Analysis 21: Comparison: ABBV-951 All Participants; Week 13 vs Baseline; Test type: Superiority — A paired-sample t-test was performed to test the change from Baseline; p < 0.001, paired-sample t-test
Statistical Analysis 22: Comparison: ABBV-951 Low Dose Subgroup; Week 26 vs Baseline; Test type: Superiority — A paired-sample t-test was performed to test the change from Baseline; p < 0.001, paired-sample t-test
Statistical Analysis 23: Comparison: ABBV-951 High Dose Subgroup; Week 26 vs Baseline; Test type: Superiority — A paired-sample t-test was performed to test the change from Baseline; p < 0.001, paired-sample t-test
Statistical Analysis 24: Comparison: ABBV-951 All Participants; Week 26 vs Baseline; Test type: Superiority — A paired-sample t-test was performed to test the change from Baseline; p < 0.001, paired-sample t-test
Statistical Analysis 25: Comparison: ABBV-951 Low Dose Subgroup; Week 39 vs Baseline; Test type: Superiority — A paired-sample t-test was performed to test the change from Baseline; p < 0.001, paired-sample t-test
Statistical Analysis 26: Comparison: ABBV-951 High Dose Subgroup; Week 39 vs Baseline; Test type: Superiority — A paired-sample t-test was performed to test the change from Baseline; p < 0.001, paired-sample t-test
Statistical Analysis 27: Comparison: ABBV-951 All Participants; Week 39 vs Baseline; Test type: Superiority — A paired-sample t-test was performed to test the change from Baseline; p < 0.001, paired-sample t-test
Statistical Analysis 28: Comparison: ABBV-951 Low Dose Subgroup; Week 52 vs Baseline; Test type: Superiority — A paired-sample t-test was performed to test the change from Baseline; p = 0.0091, paired-sample t-test
Statistical Analysis 29: Comparison: ABBV-951 High Dose Subgroup; Week 52 vs Baseline; Test type: Superiority — A paired-sample t-test was performed to test the change from Baseline; p < 0.001, paired-sample t-test
Statistical Analysis 30: Comparison: ABBV-951 All Participants; Week 52 vs Baseline; Test type: Superiority — A paired-sample t-test was performed to test the change from Baseline; p < 0.001, paired-sample t-test

56. Secondary Outcome: Movement Disorder Society-Unified Parkinson's Disease Rating Scale (MDS-UPDRS) Part III Score: Change From Baseline to End of Study
Description: The Movement Disorder Society-Unified Parkinson's Disease Rating Scale (MDS-UPDRS) is an investigator-used rating tool to follow the longitudinal course of Parkinson's Disease (PD). Part III assesses the participant's motor examination (including Hoehn and Yahr stage) with 33 questions. (The numeric score for each question is between 0-4; 0=Normal,1=Slight,2=Mild,3=Moderate,4=Severe). Part III scores range from 0 to 132, with higher scores indicating more severe symptoms of PD. Negative changes from Baseline indicate improvement.
Time Frame: Baseline, Day 2, Weeks 1, 2, 3, 4, 6, 13, 26, 39, and 52
Population: as for outcome 51
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ABBV-951 Low Dose Subgroup | ABBV-951 High Dose Subgroup | ABBV-951 All Participants
Number analyzed (Participants) | 131 | 113 | 244
units on a scale
  Day 2: number analyzed (Participants) | 120 | 102 | 222
  Day 2 | -0.6 (8.45) | -0.8 (9.20) | -0.7 (8.78)
  Week 1: number analyzed (Participants) | 119 | 106 | 225
  Week 1 | 2.0 (11.55) | 3.8 (11.00) | 2.8 (11.31)
  Week 2: number analyzed (Participants) | 117 | 94 | 211
  Week 2 | 4.1 (13.02) | 1.4 (10.93) | 2.9 (12.18)
  Week 3: number analyzed (Participants) | 107 | 96 | 203
  Week 3 | 3.9 (11.98) | 2.2 (12.07) | 3.1 (12.02)
  Week 4: number analyzed (Participants) | 107 | 93 | 200
  Week 4 | 2.7 (12.84) | 0.0 (10.97) | 1.5 (12.05)
  Week 6: number analyzed (Participants) | 104 | 89 | 193
  Week 6 | 2.4 (13.74) | -0.7 (9.58) | 0.9 (12.07)
  Week 13: number analyzed (Participants) | 89 | 70 | 159
  Week 13 | 1.4 (13.79) | -1.6 (11.82) | 0.1 (13.01)
  Week 26: number analyzed (Participants) | 75 | 64 | 139
  Week 26 | 1.4 (12.71) | 0.1 (11.61) | 0.8 (12.19)
  Week 39: number analyzed (Participants) | 75 | 55 | 130
  Week 39 | 1.9 (12.70) | 2.3 (13.26) | 2.1 (12.89)
  Week 52: number analyzed (Participants) | 75 | 58 | 133
  Week 52 | 1.8 (12.53) | 1.7 (13.02) | 1.7 (12.69)
Statistical Analysis 1: Comparison: ABBV-951 Low Dose Subgroup; Day 2 vs Baseline; Test type: Superiority — A paired-sample t-test was performed to test the change from Baseline; p = 0.4447, paired-sample t-test
Statistical Analysis 2: Comparison: ABBV-951 High Dose Subgroup; Day 2 vs Baseline; Test type: Superiority — A paired-sample t-test was performed to test the change from Baseline; p = 0.3567, paired-sample t-test
Statistical Analysis 3: Comparison: ABBV-951 All Participants; Day 2 vs Baseline; Test type: Superiority — A paired-sample t-test was performed to test the change from Baseline; p = 0.2315, paired-sample t-test
Statistical Analysis 4: Comparison: ABBV-951 Low Dose Subgroup; Week 1 vs Baseline; Test type: Superiority — A paired-sample t-test was performed to test the change from Baseline; p = 0.0667, paired-sample t-test
Statistical Analysis 5: Comparison: ABBV-951 High Dose Subgroup; Week 1 vs Baseline; Test type: Superiority — A paired-sample t-test was performed to test the change from Baseline; p < 0.001, paired-sample t-test
Statistical Analysis 6: Comparison: ABBV-951 All Participants; Week 1 vs Baseline; Test type: Superiority — A paired-sample t-test was performed to test the change from Baseline; p < 0.001, paired-sample t-test
Statistical Analysis 7: Comparison: ABBV-951 Low Dose Subgroup; Week 2 vs Baseline; Test type: Superiority — A paired-sample t-test was performed to test the change from Baseline; p < 0.001, paired-sample t-test
Statistical Analysis 8: Comparison: ABBV-951 High Dose Subgroup; Week 2 vs Baseline; Test type: Superiority — A paired-sample t-test was performed to test the change from Baseline; p = 0.2033, paired-sample t-test
Statistical Analysis 9: Comparison: ABBV-951 All Participants; Week 2 vs Baseline; Test type: Superiority — A paired-sample t-test was performed to test the change from Baseline; p < 0.001, paired-sample t-test
Statistical Analysis 10: Comparison: ABBV-951 Low Dose Subgroup; Week 3 vs Baseline; Test type: Superiority — A paired-sample t-test was performed to test the change from Baseline; p = 0.0012, paired-sample t-test
Statistical Analysis 11: Comparison: ABBV-951 High Dose Subgroup; Week 3 vs Baseline; Test type: Superiority — A paired-sample t-test was performed to test the change from Baseline; p = 0.0734, paired-sample t-test
Statistical Analysis 12: Comparison: ABBV-951 All Participants; Week 3 vs Baseline; Test type: Superiority — A paired-sample t-test was performed to test the change from Baseline; p < 0.001, paired-sample t-test
Statistical Analysis 13: Comparison: ABBV-951 Low Dose Subgroup; Week 4 vs Baseline; Test type: Superiority — A paired-sample t-test was performed to test the change from Baseline; p = 0.0304, paired-sample t-test
Statistical Analysis 14: Comparison: ABBV-951 High Dose Subgroup; Week 4 vs Baseline; Test type: Superiority — A paired-sample t-test was performed to test the change from Baseline; p > 0.999, paired-sample t-test
Statistical Analysis 15: Comparison: ABBV-951 All Participants; Week 4 vs Baseline; Test type: Superiority — A paired-sample t-test was performed to test the change from Baseline; p = 0.0891, paired-sample t-test
Statistical Analysis 16: Comparison: ABBV-951 Low Dose Subgroup; Week 6 vs Baseline; Test type: Superiority — A paired-sample t-test was performed to test the change from Baseline; p = 0.0832, paired-sample t-test
Statistical Analysis 17: Comparison: ABBV-951 High Dose Subgroup; Week 6 vs Baseline; Test type: Superiority — A paired-sample t-test was performed to test the change from Baseline; p = 0.4941, paired-sample t-test
Statistical Analysis 18: Comparison: ABBV-951 All Participants; Week 6 vs Baseline; Test type: Superiority — A paired-sample t-test was performed to test the change from Baseline; p = 0.2764, paired-sample t-test
Statistical Analysis 19: Comparison: ABBV-951 Low Dose Subgroup; Week 13 vs Baseline; Test type: Superiority — A paired-sample t-test was performed to test the change from Baseline; p = 0.3248, paired-sample t-test
Statistical Analysis 20: Comparison: ABBV-951 High Dose Subgroup; Week 13 vs Baseline; Test type: Superiority — A paired-sample t-test was performed to test the change from Baseline; p = 0.2535, paired-sample t-test
Statistical Analysis 21: Comparison: ABBV-951 All Participants; Week 13 vs Baseline; Test type: Other — A paired-sample t-test was performed to test the change from Baseline; p = 0.9274, paired-sample t-test
Statistical Analysis 22: Comparison: ABBV-951 Low Dose Subgroup; Week 26 vs Baseline; Test type: Superiority — A paired-sample t-test was performed to test the change from Baseline; p = 0.3297, paired-sample t-test
Statistical Analysis 23: Comparison: ABBV-951 High Dose Subgroup; Week 26 vs Baseline; Test type: Superiority — A paired-sample t-test was performed to test the change from Baseline; p = 0.9722, paired-sample t-test
Statistical Analysis 24: Comparison: ABBV-951 All Participants; Week 26 vs Baseline; Test type: Superiority — A paired-sample t-test was performed to test the change from Baseline; p = 0.4403, paired-sample t-test
Statistical Analysis 25: Comparison: ABBV-951 Low Dose Subgroup; Week 39 vs Baseline; Test type: Superiority — A paired-sample t-test was performed to test the change from Baseline; p = 0.1946, paired-sample t-test
Statistical Analysis 26: Comparison: ABBV-951 High Dose Subgroup; Week 39 vs Baseline; Test type: Superiority — A paired-sample t-test was performed to test the change from Baseline; p = 0.2077, paired-sample t-test
Statistical Analysis 27: Comparison: ABBV-951 All Participants; Week 39 vs Baseline; Test type: Superiority — A paired-sample t-test was performed to test the change from Baseline; p = 0.0692, paired-sample t-test
Statistical Analysis 28: Comparison: ABBV-951 Low Dose Subgroup; Week 52 vs Baseline; Test type: Superiority — A paired-sample t-test was performed to test the change from Baseline; p = 0.2276, paired-sample t-test
Statistical Analysis 29: Comparison: ABBV-951 High Dose Subgroup; Week 52 vs Baseline; Test type: Superiority — A paired-sample t-test was performed to test the change from Baseline; p = 0.3369, paired-sample t-test
Statistical Analysis 30: Comparison: ABBV-951 All Participants; Week 52 vs Baseline; Test type: Superiority — A paired-sample t-test was performed to test the change from Baseline; p = 0.1218, paired-sample t-test

57. Secondary Outcome: Movement Disorder Society-Unified Parkinson's Disease Rating Scale (MDS-UPDRS) Part IV Score: Change From Baseline to End of Study
Description: The Movement Disorder Society-Unified Parkinson's Disease Rating Scale (MDS-UPDRS) is an investigator-used rating tool to follow the longitudinal course of Parkinson's Disease (PD). Part IV assesses the participant's motor complications with 6 questions. (The numeric score for each question is between 0-4; 0=Normal,1=Slight,2=Mild,3=Moderate,4=Severe). Part IV scores range from 0 to 24, with higher scores indicating more severe symptoms of PD. Negative changes from Baseline indicate improvement.
Time Frame: Baseline, Day 2, Weeks 1, 2, 3, 4, 6, 13, 26, 39, and 52
Population: as for outcome 51
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ABBV-951 Low Dose Subgroup | ABBV-951 High Dose Subgroup | ABBV-951 All Participants
Number analyzed (Participants) | 131 | 113 | 244
units on a scale
  Day 2: number analyzed (Participants) | 117 | 101 | 218
  Day 2 | -1.8 (3.57) | -1.1 (3.45) | -1.5 (3.52)
  Week 1: number analyzed (Participants) | 117 | 105 | 222
  Week 1 | -1.7 (3.86) | -1.7 (4.10) | -1.7 (3.96)
  Week 2: number analyzed (Participants) | 115 | 93 | 208
  Week 2 | -2.5 (3.58) | -2.3 (3.56) | -2.4 (3.57)
  Week 3: number analyzed (Participants) | 102 | 96 | 198
  Week 3 | -2.1 (4.06) | -2.3 (3.74) | -2.2 (3.90)
  Week 4: number analyzed (Participants) | 106 | 94 | 200
  Week 4 | -3.0 (3.69) | -2.6 (3.78) | -2.8 (3.73)
  Week 6: number analyzed (Participants) | 101 | 89 | 190
  Week 6 | -2.6 (3.34) | -2.8 (3.90) | -2.7 (3.61)
  Week 13: number analyzed (Participants) | 89 | 77 | 166
  Week 13 | -3.7 (3.47) | -3.3 (4.04) | -3.5 (3.74)
  Week 26: number analyzed (Participants) | 77 | 69 | 146
  Week 26 | -3.5 (3.43) | -3.5 (4.12) | -3.5 (3.76)
  Week 39: number analyzed (Participants) | 73 | 59 | 132
  Week 39 | -3.5 (4.06) | -3.5 (4.11) | -3.5 (4.07)
  Week 52: number analyzed (Participants) | 72 | 58 | 130
  Week 52 | -4.1 (3.75) | -3.8 (4.71) | -3.9 (4.19)
Statistical Analysis 1: Comparison: ABBV-951 Low Dose Subgroup; Day 2 vs Baseline; Test type: Superiority — A paired-sample t-test was performed to test the change from Baseline; p < 0.001, paired-sample t-test
Statistical Analysis 2: Comparison: ABBV-951 High Dose Subgroup; Day 2 vs Baseline; Test type: Superiority — A paired-sample t-test was performed to test the change from Baseline; p = 0.0020, paired-sample t-test
Statistical Analysis 3: Comparison: ABBV-951 All Participants; Week 1 vs Baseline; Test type: Superiority — A paired-sample t-test was performed to test the change from Baseline; p < 0.001, paired-sample t-test
Statistical Analysis 4: Comparison: ABBV-951 Low Dose Subgroup; Week 1 vs Baseline; Test type: Superiority — A paired-sample t-test was performed to test the change from Baseline; p < 0.001, paired-sample t-test
Statistical Analysis 5: Comparison: ABBV-951 High Dose Subgroup; Week 1 vs Baseline; Test type: Superiority — A paired-sample t-test was performed to test the change from Baseline; p < 0.001, paired-sample t-test
Statistical Analysis 6: Comparison: ABBV-951 All Participants; Day 2 vs Baseline; Test type: Superiority — A paired-sample t-test was performed to test the change from Baseline; p < 0.001, paired-sample t-test
Statistical Analysis 7: Comparison: ABBV-951 Low Dose Subgroup; Week 2 vs Baseline; Test type: Superiority — A paired-sample t-test was performed to test the change from Baseline; p < 0.001, paired-sample t-test
Statistical Analysis 8: Comparison: ABBV-951 High Dose Subgroup; Week 2 vs Baseline; Test type: Superiority — A paired-sample t-test was performed to test the change from Baseline; p < 0.001, paired-sample t-test
Statistical Analysis 9: Comparison: ABBV-951 All Participants; Week 2 vs Baseline; Test type: Superiority — A paired-sample t-test was performed to test the change from Baseline; p < 0.001, paired-sample t-test
Statistical Analysis 10: Comparison: ABBV-951 Low Dose Subgroup; Week 3 vs Baseline; Test type: Superiority — A paired-sample t-test was performed to test the change from Baseline; p < 0.001, paired-sample t-test
Statistical Analysis 11: Comparison: ABBV-951 High Dose Subgroup; Week 3 vs Baseline; Test type: Superiority — A paired-sample t-test was performed to test the change from Baseline; p < 0.001, paired-sample t-test
Statistical Analysis 12: Comparison: ABBV-951 All Participants; Week 3 vs Baseline; Test type: Superiority — A paired-sample t-test was performed to test the change from Baseline; p < 0.001, paired-sample t-test
Statistical Analysis 13: Comparison: ABBV-951 Low Dose Subgroup; Week 4 vs Baseline; Test type: Superiority — A paired-sample t-test was performed to test the change from Baseline; p < 0.001, paired-sample t-test
Statistical Analysis 14: Comparison: ABBV-951 High Dose Subgroup; Week 4 vs Baseline; Test type: Superiority — A paired-sample t-test was performed to test the change from Baseline; p < 0.001, paired-sample t-test
Statistical Analysis 15: Comparison: ABBV-951 All Participants; Week 4 vs Baseline; Test type: Superiority — A paired-sample t-test was performed to test the change from Baseline; p < 0.001, paired-sample t-test
Statistical Analysis 16: Comparison: ABBV-951 Low Dose Subgroup; Week 6 vs Baseline; Test type: Superiority — A paired-sample t-test was performed to test the change from Baseline; p < 0.001, paired-sample t-test
Statistical Analysis 17: Comparison: ABBV-951 High Dose Subgroup; Week 6 vs Baseline; Test type: Superiority — A paired-sample t-test was performed to test the change from Baseline; p < 0.001, paired-sample t-test
Statistical Analysis 18: Comparison: ABBV-951 All Participants; Week 6 vs Baseline; Test type: Superiority — A paired-sample t-test was performed to test the change from Baseline; p < 0.001, paired-sample t-test
Statistical Analysis 19: Comparison: ABBV-951 Low Dose Subgroup; Week 13 vs Baseline; Test type: Superiority — A paired-sample t-test was performed to test the change from Baseline; p < 0.001, paired-sample t-test
Statistical Analysis 20: Comparison: ABBV-951 High Dose Subgroup; Week 13 vs Baseline; Test type: Superiority — A paired-sample t-test was performed to test the change from Baseline; p < 0.001, paired-sample t-test
Statistical Analysis 21: Comparison: ABBV-951 All Participants; Week 13 vs Baseline; Test type: Superiority — A paired-sample t-test was performed to test the change from Baseline; p < 0.001, paired-sample t-test
Statistical Analysis 22: Comparison: ABBV-951 Low Dose Subgroup; Week 26 vs Baseline; Test type: Superiority — A paired-sample t-test was performed to test the change from Baseline; p < 0.001, paired-sample t-test
Statistical Analysis 23: Comparison: ABBV-951 High Dose Subgroup; Week 26 vs Baseline; Test type: Superiority — A paired-sample t-test was performed to test the change from Baseline; p < 0.001, paired-sample t-test
Statistical Analysis 24: Comparison: ABBV-951 All Participants; Week 26 vs Baseline; Test type: Superiority — A paired-sample t-test was performed to test the change from Baseline; p < 0.001, paired-sample t-test
Statistical Analysis 25: Comparison: ABBV-951 Low Dose Subgroup; Week 39 vs Baseline; Test type: Superiority — A paired-sample t-test was performed to test the change from Baseline; p < 0.001, paired-sample t-test
Statistical Analysis 26: Comparison: ABBV-951 High Dose Subgroup; Week 39 vs Baseline; Test type: Superiority — A paired-sample t-test was performed to test the change from Baseline; p < 0.001, paired-sample t-test
Statistical Analysis 27: Comparison: ABBV-951 All Participants; Week 39 vs Baseline; Test type: Superiority — A paired-sample t-test was performed to test the change from Baseline; p < 0.001, paired-sample t-test
Statistical Analysis 28: Comparison: ABBV-951 Low Dose Subgroup; Week 52 vs Baseline; Test type: Superiority — A paired-sample t-test was performed to test the change from Baseline; p < 0.001, paired-sample t-test
Statistical Analysis 29: Comparison: ABBV-951 High Dose Subgroup; Week 52 vs Baseline; Test type: Superiority — A paired-sample t-test was performed to test the change from Baseline; p < 0.001, paired-sample t-test
Statistical Analysis 30: Comparison: ABBV-951 All Participants; Week 52 vs Baseline; Test type: Superiority — A paired-sample t-test was performed to test the change from Baseline; p < 0.001, paired-sample t-test

58. Secondary Outcome: Sleep Symptoms as Assessed by the Parkinson's Disease Sleep Scale-2 (PDSS-2) Total Score: Change From Baseline to End of Study
Description: The PDSS-2 consists of 15 questions that evaluate motor and non-motor symptoms at night and upon wakening, as well as disturbed sleep grouped into 3 domains: motor symptoms at night (5 items), Parkinson's Disease (PD) symptoms at night (5 items), and disturbed sleep (5 items). The frequency is assessed for the 15 sleep problems based on a 5-point Likert-type scale (ranging from 0 [never] to 4 [very often] with the exception of Question 1 score ranging from 0 [very often] to 4 [never]). Scores are calculated for each of the 3 domains as well as a total score. The PDSS-2 domain scores range from 0 to 20 and the total score is a sum of the 3 domains and ranges from 0 to 60. Higher scores indicate higher frequency and more severe impact of PD on sleep. Negative changes indicate improvement from Baseline.
Time Frame: Baseline, Weeks 6, 13, 26, 39, and 52
Population: as for outcome 51
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ABBV-951 Low Dose Subgroup | ABBV-951 High Dose Subgroup | ABBV-951 All Participants
Number analyzed (Participants) | 131 | 112 | 243
units on a scale
  Week 6: number analyzed (Participants) | 105 | 91 | 196
  Week 6 | -5.0 (11.39) | -7.3 (8.81) | -6.1 (10.31)
  Week 13: number analyzed (Participants) | 93 | 77 | 170
  Week 13 | -6.9 (10.76) | -8.2 (8.89) | -7.5 (9.94)
  Week 26: number analyzed (Participants) | 80 | 69 | 149
  Week 26 | -5.0 (13.06) | -8.4 (8.07) | -6.6 (11.12)
  Week 39: number analyzed (Participants) | 76 | 61 | 137
  Week 39 | -7.0 (11.19) | -7.2 (9.21) | -7.1 (10.32)
  Week 52: number analyzed (Participants) | 74 | 57 | 131
  Week 52 | -6.5 (12.34) | -8.7 (8.19) | -7.5 (10.75)
Statistical Analysis 1: Comparison: ABBV-951 Low Dose Subgroup; Week 6 vs Baseline; Test type: Superiority — A paired-sample t-test was performed to test the change from Baseline; p < 0.001, paired-sample t-test
Statistical Analysis 2: Comparison: ABBV-951 High Dose Subgroup; Week 6 vs Baseline; Test type: Superiority — A paired-sample t-test was performed to test the change from Baseline; p < 0.001, paired-sample t-test
Statistical Analysis 3: Comparison: ABBV-951 All Participants; Week 6 vs Baseline; Test type: Superiority — A paired-sample t-test was performed to test the change from Baseline; p < 0.001, paired-sample t-test
Statistical Analysis 4: Comparison: ABBV-951 Low Dose Subgroup; Week 13 vs Baseline; Test type: Superiority — A paired-sample t-test was performed to test the change from Baseline; p < 0.001, paired-sample t-test
Statistical Analysis 5: Comparison: ABBV-951 High Dose Subgroup; Week 13 vs Baseline; Test type: Superiority — A paired-sample t-test was performed to test the change from Baseline; p < 0.001, paired-sample t-test
Statistical Analysis 6: Comparison: ABBV-951 All Participants; Week 13 vs Baseline; Test type: Superiority — A paired-sample t-test was performed to test the change from Baseline; p < 0.001, paired-sample t-test
Statistical Analysis 7: Comparison: ABBV-951 Low Dose Subgroup; Week 26 vs Baseline; Test type: Superiority — A paired-sample t-test was performed to test the change from Baseline; p < 0.001, paired-sample t-test
Statistical Analysis 8: Comparison: ABBV-951 High Dose Subgroup; Week 26 vs Baseline; Test type: Superiority — A paired-sample t-test was performed to test the change from Baseline; p < 0.001, paired-sample t-test
Statistical Analysis 9: Comparison: ABBV-951 All Participants; Week 26 vs Baseline; Test type: Superiority — A paired-sample t-test was performed to test the change from Baseline; p < 0.001, paired-sample t-test
Statistical Analysis 10: Comparison: ABBV-951 Low Dose Subgroup; Week 39 vs Baseline; Test type: Other — A paired-sample t-test was performed to test the change from Baseline; p < 0.001, paired-sample t-test
Statistical Analysis 11: Comparison: ABBV-951 High Dose Subgroup; Week 39 vs Baseline; Test type: Superiority — A paired-sample t-test was performed to test the change from Baseline; p < 0.001, paired-sample t-test
Statistical Analysis 12: Comparison: ABBV-951 All Participants; Week 39 vs Baseline; Test type: Superiority — A paired-sample t-test was performed to test the change from Baseline; p < 0.001, paired-sample t-test
Statistical Analysis 13: Comparison: ABBV-951 Low Dose Subgroup; Week 52 vs Baseline; Test type: Superiority — A paired-sample t-test was performed to test the change from Baseline; p < 0.001, paired-sample t-test
Statistical Analysis 14: Comparison: ABBV-951 High Dose Subgroup; Week 52 vs Baseline; Test type: Superiority — A paired-sample t-test was performed to test the change from Baseline; p < 0.001, paired-sample t-test
Statistical Analysis 15: Comparison: ABBV-951 All Participants; Week 52 vs Baseline; Test type: Superiority — A paired-sample t-test was performed to test the change from Baseline; p < 0.001, paired-sample t-test

59. Secondary Outcome: Quality of Life Assessed by the Parkinson's Disease Questionnaire-39 Items (PDQ-39) Summary Index Score: Change From Baseline to End of Study
Description: The Parkinson's Disease Questionnaire (PDQ-39) is a disease-specific instrument designed to measure aspects of health that are relevant to participants with Parkinson's Disease (PD), and which may not be included in general health status questionnaires. Each item is scored on the following 5-point scale: 0 = never, 1 = occasionally, 2 = sometimes, 3 = often, 4 = always (or cannot do at all, if applicable). Higher scores are consistently associated with more severe symptoms of the disease such as tremors and stiffness. The results can be presented in either domain scores or as a summary index score. The full range of the PDQ-39 summary index score is from 0 (no patient-related symptoms/quality of life unaffected) to 100 (highest patient-related symptoms/low quality of life). Negative changes indicate improvement from Baseline.
Time Frame: Baseline, Weeks 6, 13, 26, 39, and 52
Population: as for outcome 51
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ABBV-951 Low Dose Subgroup | ABBV-951 High Dose Subgroup | ABBV-951 All Participants
Number analyzed (Participants) | 131 | 112 | 243
units on a scale
  Week 6: number analyzed (Participants) | 105 | 91 | 196
  Week 6 | -7.0 (14.53) | -8.4 (10.53) | -7.6 (12.81)
  Week 13: number analyzed (Participants) | 93 | 77 | 170
  Week 13 | -8.3 (15.33) | -8.2 (11.18) | -8.3 (13.57)
  Week 26: number analyzed (Participants) | 79 | 69 | 148
  Week 26 | -7.4 (13.00) | -7.1 (12.27) | -7.3 (12.62)
  Week 39: number analyzed (Participants) | 76 | 61 | 137
  Week 39 | -7.8 (13.81) | -7.5 (13.58) | -7.7 (13.66)
  Week 52: number analyzed (Participants) | 75 | 57 | 132
  Week 52 | -7.2 (14.65) | -7.2 (12.35) | -7.2 (13.65)
Statistical Analysis 1: Comparison: ABBV-951 Low Dose Subgroup; Week 6 vs Baseline; Test type: Superiority — A paired-sample t-test was performed to test the change from Baseline; p < 0.001, paired-sample t-test
Statistical Analysis 2: Comparison: ABBV-951 High Dose Subgroup; Week 6 vs Baseline; Test type: Superiority — A paired-sample t-test was performed to test the change from Baseline; p < 0.001, paired-sample t-test
Statistical Analysis 3: Comparison: ABBV-951 All Participants; Week 6 vs Baseline; Test type: Superiority — A paired-sample t-test was performed to test the change from Baseline; p < 0.001, paired-sample t-test
Statistical Analysis 4: Comparison: ABBV-951 Low Dose Subgroup; Week 13 vs Baseline; Test type: Superiority — A paired-sample t-test was performed to test the change from Baseline; p < 0.001, paired-sample t-test
Statistical Analysis 5: Comparison: ABBV-951 High Dose Subgroup; Week 13 vs Baseline; Test type: Superiority — A paired-sample t-test was performed to test the change from Baseline; p < 0.001, paired-sample t-test
Statistical Analysis 6: Comparison: ABBV-951 All Participants; Week 13 vs Baseline; Test type: Superiority — A paired-sample t-test was performed to test the change from Baseline; p < 0.001, paired-sample t-test
Statistical Analysis 7: Comparison: ABBV-951 Low Dose Subgroup; Week 26 vs Baseline; Test type: Superiority — A paired-sample t-test was performed to test the change from Baseline; p < 0.001, paired-sample t-test
Statistical Analysis 8: Comparison: ABBV-951 High Dose Subgroup; Week 26 vs Baseline; Test type: Superiority — A paired-sample t-test was performed to test the change from Baseline; p < 0.001, paired-sample t-test
Statistical Analysis 9: Comparison: ABBV-951 All Participants; Week 26 vs Baseline; Test type: Superiority — A paired-sample t-test was performed to test the change from Baseline; p < 0.001, paired-sample t-test
Statistical Analysis 10: Comparison: ABBV-951 Low Dose Subgroup; Week 39 vs Baseline; Test type: Superiority — A paired-sample t-test was performed to test the change from Baseline; p < 0.001, paired-sample t-test
Statistical Analysis 11: Comparison: ABBV-951 High Dose Subgroup; Week 39 vs Baseline; Test type: Superiority — A paired-sample t-test was performed to test the change from Baseline; p < 0.001, paired-sample t-test
Statistical Analysis 12: Comparison: ABBV-951 All Participants; Week 39 vs Baseline; Test type: Superiority — A paired-sample t-test was performed to test the change from Baseline; p < 0.001, paired-sample t-test
Statistical Analysis 13: Comparison: ABBV-951 Low Dose Subgroup; Week 52 vs Baseline; Test type: Superiority — A paired-sample t-test was performed to test the change from Baseline; p < 0.001, paired-sample t-test
Statistical Analysis 14: Comparison: ABBV-951 High Dose Subgroup; Week 52 vs Baseline; Test type: Other — A paired-sample t-test was performed to test the change from Baseline; p < 0.001, paired-sample t-test
Statistical Analysis 15: Comparison: ABBV-951 All Participants; Week 52 vs Baseline; Test type: Superiority — A paired-sample t-test was performed to test the change from Baseline; p < 0.001, paired-sample t-test

60. Secondary Outcome: The EuroQol 5-Dimension Questionnaire (EQ-5D-5L) Quality of Life Summary Index: Change From Baseline to End of Study
Description: The EuroQol 5-dimension questionnaire (EQ-5D-5L) is a standardized non-disease specific instrument for describing and valuing health-related quality of life. The EQ-5D-5L descriptive system comprises 5 dimensions of health (mobility, self -care, usual activities, pain/discomfort, and anxiety/depression) to describe the participant's current health state. Each dimension comprises 5 levels with corresponding numeric scores, where 1 indicates no problems, and 5 indicates extreme problems. The health status is converted to an index value using the country-specific weighted scoring algorithm for the United States (US). The summary index value for the US ranges from a worst score of -0.109 to a best score of 1. An increase in the EQ-5D-5L total score indicates improvement.
Time Frame: Baseline, Weeks 6, 13, 26, 39, and 52
Population: as for outcome 51
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ABBV-951 Low Dose Subgroup | ABBV-951 High Dose Subgroup | ABBV-951 All Participants
Number analyzed (Participants) | 125 | 104 | 229
units on a scale
  Week 6: number analyzed (Participants) | 93 | 82 | 175
  Week 6 | 0.060 (0.1921) | 0.113 (0.1780) | 0.085 (0.1870)
  Week 13: number analyzed (Participants) | 80 | 66 | 146
  Week 13 | 0.064 (0.2153) | 0.122 (0.1984) | 0.090 (0.2092)
  Week 26: number analyzed (Participants) | 70 | 58 | 128
  Week 26 | 0.074 (0.1771) | 0.122 (0.1803) | 0.096 (0.1795)
  Week 39: number analyzed (Participants) | 72 | 49 | 121
  Week 39 | 0.075 (0.1842) | 0.129 (0.1995) | 0.097 (0.1916)
  Week 52: number analyzed (Participants) | 70 | 52 | 122
  Week 52 | 0.076 (0.2062) | 0.126 (0.2213) | 0.097 (0.2134)
Statistical Analysis 1: Comparison: ABBV-951 Low Dose Subgroup; Week 6 vs Baseline; Test type: Superiority — A paired-sample t-test was performed to test the change from Baseline; p = 0.0035, paired-sample t-test
Statistical Analysis 2: Comparison: ABBV-951 High Dose Subgroup; Week 6 vs Baseline; Test type: Superiority — A paired-sample t-test was performed to test the change from Baseline; p < 0.001, paired-sample t-test
Statistical Analysis 3: Comparison: ABBV-951 All Participants; Week 6 vs Baseline; Test type: Superiority — A paired-sample t-test was performed to test the change from Baseline; p < 0.001, paired-sample t-test
Statistical Analysis 4: Comparison: ABBV-951 Low Dose Subgroup; Week 13 vs Baseline; Test type: Superiority — A paired-sample t-test was performed to test the change from Baseline; p = 0.0098, paired-sample t-test
Statistical Analysis 5: Comparison: ABBV-951 High Dose Subgroup; Week 13 vs Baseline; Test type: Superiority — A paired-sample t-test was performed to test the change from Baseline; p < 0.001, paired-sample t-test
Statistical Analysis 6: Comparison: ABBV-951 All Participants; Week 13 vs Baseline; Test type: Superiority — A paired-sample t-test was performed to test the change from Baseline; p < 0.001, paired-sample t-test
Statistical Analysis 7: Comparison: ABBV-951 Low Dose Subgroup; Week 26 vs Baseline; Test type: Superiority — A paired-sample t-test was performed to test the change from Baseline; p < 0.001, paired-sample t-test
Statistical Analysis 8: Comparison: ABBV-951 High Dose Subgroup; Week 26 vs Baseline; Test type: Superiority — A paired-sample t-test was performed to test the change from Baseline; p < 0.001, paired-sample t-test
Statistical Analysis 9: Comparison: ABBV-951 All Participants; Week 26 vs Baseline; Test type: Superiority — A paired-sample t-test was performed to test the change from Baseline; p < 0.001, paired-sample t-test
Statistical Analysis 10: Comparison: ABBV-951 Low Dose Subgroup; Week 39 vs Baseline; Test type: Superiority — A paired-sample t-test was performed to test the change from Baseline; p < 0.001, paired-sample t-test
Statistical Analysis 11: Comparison: ABBV-951 High Dose Subgroup; Week 39 vs Baseline; Test type: Superiority — A paired-sample t-test was performed to test the change from Baseline; p < 0.001, paired-sample t-test
Statistical Analysis 12: Comparison: ABBV-951 All Participants; Week 39 vs Baseline; Test type: Superiority — A paired-sample t-test was performed to test the change from Baseline; p < 0.001, paired-sample t-test
Statistical Analysis 13: Comparison: ABBV-951 Low Dose Subgroup; Week 52 vs Baseline; Test type: Superiority — A paired-sample t-test was performed to test the change from Baseline; p = 0.0030, paired-sample t-test
Statistical Analysis 14: Comparison: ABBV-951 High Dose Subgroup; Week 52 vs Baseline; Test type: Superiority — A paired-sample t-test was performed to test the change from Baseline; p < 0.001, paired-sample t-test
Statistical Analysis 15: Comparison: ABBV-951 All Participants; Week 52 vs Baseline; Test type: Superiority — A paired-sample t-test was performed to test the change from Baseline; p < 0.001, paired-sample t-test

ADVERSE EVENTS:
Time Frame: All-cause mortality is reported from enrollment to end of study; median time on follow-up was 367.0 days for the ABBV-951 Low Dose Subgroup, the ABBV-951 High Dose Subgroup, and the ABBV-951 All Participants group. TEAEs and SAEs were collected from first dose of study drug until 30 days after the last infusion; mean time on treatment was 244.9 days for the ABBV-951 Low Dose Subgroup, 240.6 days for the ABBV-951 High Dose Subgroup, and 242.9 days for the ABBV-951 All Participants group.
Arm/Group | ABBV-951 Low Dose Subgroup | ABBV-951 High Dose Subgroup | ABBV-951 All Participants
All-Cause Mortality (participants affected / at risk) | 0/131 | 5/113 | 5/244
Serious Adverse Events (participants affected / at risk) | 32/131 | 31/113 | 63/244
Other Adverse Events (participants affected / at risk) | 111/131 | 107/113 | 218/244
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ABBV-951 Low Dose Subgroup (N=131) | ABBV-951 High Dose Subgroup (N=113) | ABBV-951 All Participants (N=244)
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
ATRIAL FIBRILLATION (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1)
CARDIAC ARREST (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
CARDIO-RESPIRATORY ARREST (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1)
CORONARY ARTERY DISEASE (Cardiac disorders) | 1 (1) | 1 (1) | 2 (2)
PERIORBITAL PAIN (Eye disorders) | 0 (0) | 1 (1) | 1 (1)
PERIORBITAL SWELLING (Eye disorders) | 0 (0) | 1 (1) | 1 (1)
COLITIS ISCHAEMIC (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
INTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
ASTHENIA (General disorders) | 1 (1) | 0 (0) | 1 (1)
CHEST DISCOMFORT (General disorders) | 0 (0) | 1 (1) | 1 (1)
CHEST PAIN (General disorders) | 1 (1) | 0 (0) | 1 (1)
HYPOTHERMIA (General disorders) | 1 (1) | 0 (0) | 1 (1)
INFUSION SITE HAEMATOMA (General disorders) | 0 (0) | 1 (1) | 1 (1)
INFUSION SITE INJURY (General disorders) | 0 (0) | 1 (1) | 1 (1)
ABSCESS LIMB (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
COVID-19 (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
CELLULITIS (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
INFUSION SITE ABSCESS (Infections and infestations) | 5 (5) | 3 (5) | 8 (10)
INFUSION SITE CELLULITIS (Infections and infestations) | 4 (4) | 6 (6) | 10 (10)
INFUSION SITE INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
PAROTID ABSCESS (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
PNEUMONIA (Infections and infestations) | 2 (2) | 1 (2) | 3 (4)
SEPSIS (Infections and infestations) | 3 (3) | 0 (0) | 3 (3)
SEPTIC SHOCK (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
URINARY TRACT INFECTION (Infections and infestations) | 2 (2) | 2 (2) | 4 (4)
FACE INJURY (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
FALL (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 2 (2)
SUBDURAL HAEMATOMA (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
BLOOD SODIUM DECREASED (Investigations) | 1 (1) | 0 (0) | 1 (1)
DEHYDRATION (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1)
HYPOKALAEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1)
HYPONATRAEMIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1)
ARTHRITIS REACTIVE (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
RHABDOMYOLYSIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
SACROILIAC JOINT DYSFUNCTION (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
RECTAL ADENOCARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1)
CEREBRAL MASS EFFECT (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
COGNITIVE DISORDER (Nervous system disorders) | 1 (1) | 1 (1) | 2 (2)
DIZZINESS (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
DYSARTHRIA (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
DYSTONIA (Nervous system disorders) | 0 (0) | 2 (3) | 2 (3)
GENERALISED TONIC-CLONIC SEIZURE (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
HEMIANAESTHESIA (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
HEMIPARESIS (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
LOSS OF CONSCIOUSNESS (Nervous system disorders) | 1 (1) | 1 (1) | 2 (2)
LUMBOSACRAL RADICULOPATHY (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
ON AND OFF PHENOMENON (Nervous system disorders) | 1 (2) | 0 (0) | 1 (2)
PARAESTHESIA (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
PARKINSON'S DISEASE (Nervous system disorders) | 5 (6) | 1 (1) | 6 (7)
PARKINSONISM (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
PSYCHOGENIC SEIZURE (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
ANXIETY (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1)
CONFUSIONAL STATE (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1)
DELIRIUM (Psychiatric disorders) | 1 (1) | 1 (1) | 2 (2)
DELUSION (Psychiatric disorders) | 1 (1) | 1 (1) | 2 (2)
DELUSIONAL DISORDER, UNSPECIFIED TYPE (Psychiatric disorders) | 0 (0) | 1 (1) | 1 (1)
DOPAMINE DYSREGULATION SYNDROME (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1)
HALLUCINATION (Psychiatric disorders) | 6 (6) | 1 (1) | 7 (7)
PSYCHOTIC DISORDER (Psychiatric disorders) | 4 (5) | 2 (2) | 6 (7)
SUICIDE ATTEMPT (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1)
BRONCHIECTASIS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
HYPERVENTILATION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
HAEMATOMA (Vascular disorders) | 0 (0) | 1 (1) | 1 (1)
HAEMORRHAGE (Vascular disorders) | 0 (0) | 1 (1) | 1 (1)
ORTHOSTATIC HYPOTENSION (Vascular disorders) | 1 (1) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ABBV-951 Low Dose Subgroup (N=131) | ABBV-951 High Dose Subgroup (N=113) | ABBV-951 All Participants (N=244)
CONSTIPATION (Gastrointestinal disorders) | 8 (8) | 12 (12) | 20 (20)
NAUSEA (Gastrointestinal disorders) | 8 (11) | 11 (13) | 19 (24)
INFUSION SITE BRUISING (General disorders) | 10 (15) | 8 (15) | 18 (30)
INFUSION SITE ERYTHEMA (General disorders) | 64 (175) | 63 (168) | 127 (343)
INFUSION SITE EXTRAVASATION (General disorders) | 8 (10) | 12 (15) | 20 (25)
INFUSION SITE HAEMATOMA (General disorders) | 10 (10) | 7 (12) | 17 (22)
INFUSION SITE INFLAMMATION (General disorders) | 3 (3) | 6 (9) | 9 (12)
INFUSION SITE NODULE (General disorders) | 36 (65) | 34 (58) | 70 (123)
INFUSION SITE OEDEMA (General disorders) | 19 (78) | 28 (45) | 47 (123)
INFUSION SITE PAIN (General disorders) | 18 (41) | 20 (27) | 38 (68)
INFUSION SITE PAPULE (General disorders) | 7 (8) | 11 (18) | 18 (26)
INFUSION SITE REACTION (General disorders) | 13 (26) | 17 (36) | 30 (62)
INJECTION SITE ERYTHEMA (General disorders) | 6 (22) | 8 (14) | 14 (36)
INJECTION SITE NODULE (General disorders) | 3 (15) | 6 (8) | 9 (23)
INJECTION SITE PAIN (General disorders) | 2 (2) | 6 (6) | 8 (8)
INFUSION SITE ABSCESS (Infections and infestations) | 9 (9) | 10 (12) | 19 (21)
INFUSION SITE CELLULITIS (Infections and infestations) | 25 (33) | 21 (31) | 46 (64)
INFUSION SITE INFECTION (Infections and infestations) | 7 (8) | 10 (16) | 17 (24)
URINARY TRACT INFECTION (Infections and infestations) | 6 (7) | 9 (14) | 15 (21)
CONTUSION (Injury, poisoning and procedural complications) | 2 (3) | 6 (9) | 8 (12)
FALL (Injury, poisoning and procedural complications) | 16 (42) | 23 (35) | 39 (77)
SKIN LACERATION (Injury, poisoning and procedural complications) | 1 (1) | 6 (6) | 7 (7)
VITAMIN B6 DECREASED (Investigations) | 5 (5) | 6 (6) | 11 (11)
WEIGHT DECREASED (Investigations) | 10 (10) | 14 (14) | 24 (24)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 8 (8) | 5 (6) | 13 (14)
DIZZINESS (Nervous system disorders) | 14 (18) | 10 (10) | 24 (28)
DYSKINESIA (Nervous system disorders) | 12 (20) | 6 (7) | 18 (27)
HEADACHE (Nervous system disorders) | 7 (7) | 7 (10) | 14 (17)
PARKINSON'S DISEASE (Nervous system disorders) | 7 (8) | 4 (4) | 11 (12)
SOMNOLENCE (Nervous system disorders) | 9 (11) | 3 (3) | 12 (14)
ANXIETY (Psychiatric disorders) | 10 (12) | 18 (22) | 28 (34)
DELUSION (Psychiatric disorders) | 7 (8) | 1 (1) | 8 (9)
HALLUCINATION (Psychiatric disorders) | 14 (22) | 21 (27) | 35 (49)
HALLUCINATION, VISUAL (Psychiatric disorders) | 10 (14) | 5 (6) | 15 (20)
INSOMNIA (Psychiatric disorders) | 9 (9) | 9 (9) | 18 (18)
ORTHOSTATIC HYPOTENSION (Vascular disorders) | 6 (6) | 6 (7) | 12 (13)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (2):
  • Study Protocol (2021-02-11): https://cdn.clinicaltrials.gov/large-docs/67/NCT03781167/Prot_000.pdf
  • Statistical Analysis Plan (2021-03-10): https://cdn.clinicaltrials.gov/large-docs/67/NCT03781167/SAP_001.pdf